# CITY OF HOPE NATIONAL MEDICAL CENTER 1500 E. Duarte Road Duarte, CA 91010

#### **Division of Hematology and Hematopoietic Cell Transplantation**

TITLE: Phase II Study of IV Busulfan Combined with 12 Gy of Fractionated Total Body Irradiation (FTBI) and

Etoposide (VP16) as a Preparative Regimen for Allogeneic Hematopoietic Stem Cell (HSC)

Transplantation for Patients with Advanced Hematological Malignancies

CITY OF HOPE PROTOCOL NUMBER/VERSION NUMBER: IRB# 99041 PROTOCOL DATE: 04/20/2004

DATE(S) AMENDMENT(S)/REVISION(S)

| Amendment 1 | 08/28/00 | Version 01 |
|------------------------------|------------------------------|-------------|
| Amendment 2 | 11/08/01 | Version 02 |
| Amendment 3 | 03/11/02 | Version 03 |
| Amendment 4 | 06/13/02 | Version 04 |
| Amendment 5 | 08/12/02 | Version 05 |
| (Consent form change | 10/16/02 | Version 05) |
| Amendment 6 | 11/18/02 | Version 06 |
| Amendment 7 | 04/20/04 | Version 07 |
| Amendment 8 | 09/28/17 | Version 08 |
| Amendment 9 | 07/26/19 | Version 09 |
| Amendment 10 at Continuation | 07/01/20 | Version 10 |
| Amendment 11 at Continuation | Protocol Dated 04/20/04 (TP) | Packet 11 |

**HISTOLOGY**: Advanced Hematological Malignancies

**STAGE**: Advanced **MODALITY:** Allogeneic BMT

TYPE: Phase II

**Principal Investigator at COH:** Anthony Stein, M.D.

**Collaborating Investigator(s):** Stephen J. Forman, M.D.

Joyce Niland, Ph.D.

**Participating Clinicians:** 

Amrita Krishnan, M.D.

Leslie Popplewell, M.D. Eileen Smith, M.D. Jasmine Zain, M.D.

Ricardo Spielberger, M.D.

Department of Medical Oncology Kim Margolin, M.D.

Tim Synold, Ph.D.

Department of Pediatric/BMT Joseph Rosenthal, M.D. Department of Radiation Oncology Nayana Vora, M.D.

City of Hope Samaritan Bone Marrow Joseph C. Alvarnas, M.D.

**Transplantation Program** 

IRB # 99041 04/20/04

Packet: 11

#### **SCHEMA**

Rev. 11/8/01



### TABLE OF CONTENTS

| 1.0 | Objec | tives | 3 |
|------|----------|--------------------------------------------------|----|
| 2.0 | Backg | ground & Hypothesis | 3 |
| 3.0 | Drug | Information | 4 |
| 4.0 | Stagir | ng Criteria | 9 |
| 5.0 | Eligibi | ility Criteria | 10 |
| 6.0 | Treatr | ment Plan | 11 |
| 7.0 | Toxici | ties to be Monitored and Dose Modifications | 15 |
| 8.0 | Toxici | ty Grading Scale | 16 |
| 9.0 | Study | Calendar | 16 |
| 10.0 | Criteri | ia for Evaluation and Definition | 16 |
| 11.0 | Criteri | ia for Removal from Study | 17 |
| 12.0 | | tical Considerations | 17 |
| 13.0 | | en and Minorities Guidelines | 18 |
| 14.0 | | lines for Reporting Adverse Events | 18 |
| 15.0 | Refer | ences | 19 |
| Appe | ndix l | IV Busulfan Kinetics Form | 22 |
| Appe | ndix II | Fractionated Total Body Irradiation Schema | 23 |
| Appe | ndix III | | 24 |
| Appe | ndix IV | Acute GVHD staging and grading table | 25 |
| | | Grading of Chronic GVHD | 26 |
| | | Study Calendar | 27 |
| | | Common Toxicity Criteria (Version 2.0) | 28 |
| | | IIGuidelines for reporting of adverse events | 66 |
| | | Eligibility Checklist | 67 |
| Appe | ndix X | Time points to grade toxicities and collect data | 68 |

#### 1.0OBJECTIVES

1.1 To determine the efficacy of intravenous busulfan, dose targeted to achieve AUC of 700-900 combined with fractionated total body irradiation and VP16 as a preparative regimen for marrow transplantation from an HLA-identical sibling in patients with advanced hematological malignancies (AML or ALL) beyond 2<sup>nd</sup> remission, induction failure, in relapse, chronic myelogenous leukemia in blast crisis and myelodysplasia (RAEB and RAEBIT).

Rev. 6/13/02

- 1.2 To determine the efficacy of this regimen in patients with AML in first remission with unfavorable cytogenetics.
- 1.3 To evaluate the early and late toxicities of this regimen.

#### 2.0 BACKGROUND AND HYPOTHESIS

During the last 20 years clinical bone marrow transplantation from a histocompatible sibling donor has evolved into an important treatment modality for patients with acute lymphoblastic leukemia, acute myelogenous leukemia and chronic myelogenous leukemia. If the transplant procedure is performed in first complete remission of acute leukemia or during chronic phase or chronic myelogenous leukemia, approximately 50-70% of patients become disease free long-term survivors. (1-8) In contrast, the chances for an ultimately successful outcome of bone marrow transplantation drops to 10-40% if this is performed during second or subsequent complete remission, during relapse of acute leukemias, or while patients with chronic myelogenous leukemia are in accelerated or blast phase of this disease. In the latter group of patients the probability of leukemic relapse is in the range of 40-70%. (9-16) Many transplant centers have performed several phase I-II trials of preparative regimens using alternative chemotherapeutic agents or methods of administering TBI. Some of these studies suggest a decrease in the post-transplant relapse rate that are often associated with increased transplant related morbidity and mortality from regimen related toxicity. (17-20) At the City of Hope a phase I/II trial was conducted in 1986 to determine the efficacy of substituting etoposide (VP-16) for cyclophosphamide in combination with fractionated total body irradiation (FTBI). This trial was done in 33 patients with acute leukemia beyond first remission, and resulted in a 43% longterm disease free survivorship. Despite this improved survival compared to previous studies there still is significant relapse rate, particularly in patients with advanced leukemia. This regimen has subsequently been utilized to treat 100 patients with acute leukemia in remission. There was only one case of fatal venoocclusive disease; otherwise the regimen was well tolerated. (21) combining busulfan and cyclophosphamide as a preparative regimen for patients with advanced hematological malignancies have been reported to result in similar or superior outcomes when compared with standard cyclophosphamide and TBI regimens, suggesting that busulfan has important anti-leukemic effects. randomized Southwest Oncology Group study (SWOG) comparing busulfan, cyclosphophamide with FTBI VP-16 showed 20% disease free survival for patients transplanted with advanced leukemia. (22) At City of Hope a phase I study was conducted utilizing escalating doses busulfan in combination with fixed doses of FTBI and VP-16 in an attempt to decrease the relapse rate in those patients transplanted for advanced hematological malignancies. The rationale behind the study was that we combined three non-cross resistant anti-leukemic agents with non-overlapping extramedullary toxicities. An in vitro synergy has been demonstrated between busulfan/VP-16 and busulfan/VP-16 has been proven to be an effective regimen for relapsed leukemia and for ABMT for AML in first and second remission. The dose limiting toxicity occurred at 12mg/kg the MTD was defined at 11mg/kg. At this dose level median first dose AUC for these patients was 892μM\*min (460-1267). With a median follow-up of 11.5 months, the disease-free survival is 32%, and the probability of relapse is 40%. The only variable predictive of a disease-free survival and relapse was the busulfan dose of 7-8 mg/kg. In this phase I study there was a wide variability of the AUC of busulfan due to the variability of absorption of oral busulfan. An AUC of 700-950 showed a trend to a decreased relapse rate and improved disease free survival.

A phase II study utilizing IV busulfan was conducted at City of Hope which has resulted in FDA approval of IV busulfan and it is proposed to substitute IV busulfan which has been shown to have more predictable pharmacokinetic properties than the oral preparation resulting in a better toxicity profile. (25,26,27)

Rev. 6/13/02

\*Patients with AML in first complete remission (CR1) with unfavorable cytogenetics have a relapse rate of 40% with our current transplant regimen consisting of fractionated radiation and etoposide. We propose to use this new preparative regimen to see if it can improve the DFS and relapse rate for this subset of patients with AML in first CR.

#### 3.0 DRUG INFORMATION

#### 3.1 Busulfan (Myleran)

- 3.11 Mechanism of Action: Busulfan is a bifunctional alkylating agent. In aqueous media, busulfan hydrolyses to produce reactive carbonium ions that can alkylate DNA.
- 3.12 Formulation and stability: Busulfan injection is a sterile, pyrogen-free solution provided in a mixture of dimethylacetamide (DMA) and polyethlyeneglycol 400 (PEG 400). It is supplied in 10-ml single use ampules at a concentration of 6-mg Busulfan per ml. Each ampule contains 60mg of Busulfan in 3.3 ml of DMA and 6.7 ml of PEG 400. When diluted in normal saline or D5W to a concentration of 0.5mg/mL, the resulting solution must be administered within eight (8) hours of preparation; including the 2 hours of infusion of the drug.

Stable at 4° C for at least twelve months. Ampules should be stored refrigerated at 2-8° C. Do not freeze. Ampules may be stored for up to seven days at room temperature.

Solution preparation: prepare the Busulfan solution as follows: Use sterile, non-pyrogenic, disposable containers, syringes, needles, stopcocks, and transfer tubing, etc. Calculate the amount of drug to be administrated based on the dosage and the patient's body weight.

Prepare a solution of 0.9% sodium chloride injection USP (normal saline) calculated Busulfan dose in ml from the step above.

Break off the top of the ampule and remove the calculated volume of Busulfan from the container by using a syringe fitted with a filter needle or equivalent. Transfer the contents of the syringe into the calculated amount of either normal saline or D5W making sure that the drug flows into and through the solution. Mix by inverting the bag.

- 3.13 Administration: Each dose of the drug will be given by slow central intravenous infusion over 2 hours. Caution: Do not administer as an intravenous push or bolus.
- 3.14 Supplier: This drug is commercially available; manufactured by Orphan Medical Inc.
- 3.15 Toxicity: Toxicity from busulfan includes:
  - a). Severe bone marrow hypoplasia, which would be fatal without administration of bone marrow, stem cells.
  - b). Nausea and vomiting which can be decreased by the use of sedation and anti-emetics.
  - c). Stomatitis and diarrhea which can be treated symptomatically with fluid replacement and atropine or diphenoxylate H C1.
  - d). Pulmonary fibrosis characterized by delayed onset of cough, shortness of breath and low-grade fever.
  - e). Hepatic damage, which can occur in combination with cytoxan or as a single agent and can result in significant hepatic toxicity which, can be fatal.
  - f). Temporary hyperpigmentation of the skin and nail bed changes.
  - g). Grand mal seizures which can be prevented by the prophylactic administration of Dilantin.
- 3.2 VP-16 (VP-16-213) (Etoposide) (Vepesid)
  - 3.21 <u>Chemistry</u>: VP-16 is a semi-synthetic podophyllotoxin derivative from the plant podophyllum pletatum, has anti-neoplastic properties in experimental animals and in man. The empiric formula  $C_{29}$   $H_{32}$   $0_{13}$  has a molecular weight of 588.
  - Mechanism of Action: The epipodophyllotoxin exert phase-specific spindle poison activity with metaphase arrest, but in contrast to the vinca alkaloids, have an additional activity of inhibiting cells from entering mitosis. Suppression of tritiated thymidine, uridine, and leucine incorporation in human cells in tissue culture suggest effects against DNA, RNA and protein synthesis.
  - 3.23 <u>Animal Tumor Data</u>: Significant anti-tumor effect has been demonstrated in L-1210, mouse sarcoma 37 and 180, Walker carcinosarcoma and Erlich ascites tumor. With the L 1210 system,

activity was schedule-dependent, having greater effect with a twice a week administration than with daily dosing or the administration of single large doses. The drug is active given intraperitoneally or orally in L 1210. No effect was demonstrated intracerebrally inoculated L 1210.

- Animal Toxicology: The predominant toxicities of VP-16 in animal studies involve the hematopoietic system, with toxicity to the liver and GI tract occurring only at doses producing profound myelosuppression. Anemia, leukopenia, and lymphoid involution occur in mice, rats and monkeys. Acute toxicity investigations have been complicated by the toxicity of the solvent system. The LD-50 of the solvent plus drug approached that of the solvent alone. Immuno-suppressive effects occur with an inhibition of antibody production in mice and monkeys, and prevention of experimental allergic encephalomyelitis in rats (cell mediated immunity).
- 3.25 <u>Human Toxicology</u>: Reversible myelotoxicity has been uniformly observed to be the major toxicity of VP-16 and to represent the only clinically significant side effect. Following a single IV injection, peak myelotoxicity occurs at 7 to 9 days. Following daily IV injections for 5 to 7 days, myelotoxicity is maximal between 12 to 16 days from the initiation of therapy. Bone marrow suppression is mainly manifested as granulocytopenia with thrombocytopenia and anemia occurring to a lesser extent. Transient, modest nausea, usually without vomiting, is common. Occasional alopecia is reported. VP-16 does not produce stomatitis, phlebitis, neurotoxicity, hepato-toxicity or nephro-toxicity. Hypotension and anaphylaxis are occasional side effects. Hypotension can be managed by infusing the drug over at least a 30 minute period. Occasionally, fever may be a result of VP-16 administration.
- 3.26 Pharmaceutical Data: Formulation: 100 mg of VP-16 is supplied as 5 ml of solution in <u>clear</u> ampules for injection. Each ampule also contains anhydrous citric acid 10 mg, benzylalcohol 150 mg, polysorbate 80 purified 400 mg, polyethylene glycol and absolute alcohol. The contents of the ampule are non-aqueous and <u>must be diluted</u> with 20 to 50 volumes of <u>sodium chloride injection USP</u>. The time before precipitation depends on concentration.

| <u>Dilution</u> | <u>Time</u> |
|-----------------|--------------------|
| 1:20<br>1:50 | 30 minutes 3 hours |
| 1:100 | 6 hours |

3.27 <u>Storage and stability</u>: The drug is available as a box of 10 ampules that are stored at room temperature. Each ampule should be kept in the box to protect it from light. VP-16 is less stable in 5% Dextrose injection and precipitation is reported. VP-16 has a <u>minimum infusion time of 30 minutes</u> to reduce hypotension.

3.28 <u>Supplier</u>: VP-16 is commercially available.

#### 3.3 Cyclosporine:

- 3.31 <u>Mechanism of Action</u>: Cyclosporine is an immunosuppressant used to prevent the rejection of transplanted kidneys, hearts and livers. It is also effective in treating bone marrow recipients with acute graft vs host disease. The drug inhibits T lymphocyte function with minimal activity against B cells.
- 3.32 <u>Human Toxicology:</u> Nephrotoxicity is the most frequent side effect of cyclosporine. Other frequently observed side effects include hypertension, hirsutism, tremors, paresthesias, hepato-toxicity, hypomagnesemia and hyperkalemia. Transient gastrointestinal symptoms have also occurred, to include anorexia, nausea and ileus. The drug has demonstrated a relative lack of myelotoxicity.
- 3.33 Pharmaceutical Data: Formulation: Cyclosporine is available for oral and intravenous administration. Cyclosporine is an olive oil solution supplied in 50 ml bottles containing 100 mg/ml. The intravenous solution is available as 5 ml ampules containing 50 mg/ml. Cyclosporine is also available as 25mg and 100mg capsules.
- 3.34 <u>Storage and Stability</u>: The oral solution of cyclosporine should be stored and dispensed in the original container at temperatures below 86°F and should be used within two months after opening bottle. Do not store in the refrigerator. The intravenous solution should be stored at temperatures below 86°F and protected from light.
- 3.35 <u>Administration:</u> The oral solution may be mixed with whole milk, chocolate milk or fruit juice to mask the taste and should be taken immediately after mixing. Cyclosporine should be administered intravenously over 2 to 6 hours. Longer infusion times are acceptable and sometimes better tolerated. The contents of the ampule should be diluted with 50-250 ml of 0.9% sodium chloride injection or 5% dextrose injection.
  - 3.36 Supplier: This drug is commercially available.

#### 3.4 Methotrexate

- 3.41 <u>Chemistry</u>: Methotrexate is a well known antimetabolite which has been intensively studied.
- 3.42 <u>Biochemistry</u>: As a folic acid analog, methotrexate is considered to act as an inhibitor or dihydrofolate reductase to which it tightly binds.
- 3.43 <u>Human Pharmacology</u>: Methotrexate is well absorbed in low doses from the gastrointestinal tract and is well absorbed when given intramuscularly. Large doses are completely absorbed when given

orally. About 40-50% of small doses and about 90% of large doses are excreted unchanged in the urine within eight hours. Toxicity is directly related to the duration of blood levels and thus, renal insufficiency can significantly increase toxicity. In man, there is insignificant metabolism of methotrexate.

- 3.44 <u>Human Toxicity</u>: Human toxicity includes myelosuppression, mucositis, nausea and abdominal discomfort, generalized malaise, rashes, photosensitization, decreased renal function, fetal death, hepatic toxicity and pulmonary toxicity (methotrexate lung).
- 3.45 Pharmaceutical Data: Formulation; 50mg vials containing 25mg/cc.
- 3.46 Storage: Room temperature.
- 3.47 <u>Administration:</u> In this study, administered intravenously.
- 3.48 <u>Supplier:</u> Methotrexate is commercially available for purchase by the third party.

#### 4.0 STAGING CRITERIA:

4.1 Definition of Disease Stages of Chronic Myelogenous Leukemia

#### Chronic Phase

- 1. No significant symptoms which are not readily controlled by conventional doses of hydroxyurea or busulfan.
- 2. None of the features of accelerated phase or blastic phase. (Note: Granulocytic hyperplasia and the Philadelphia chromosome may be present in the bone marrow).

#### <u>Accelerated Phase</u> (any one or more of the following criteria)

- 1. WBC difficult to control with conventional use of busulfan/hydroxyurea in terms of doses required or shortening of intervals between courses.
- Rapid doubling of WBC (< 5 days).</li>
- 3. > 10% blasts in blood or marrow.
- 4. > 20% blasts plus promyelocytes in blood or marrow.
- 5. > 20% basophils plus eosinophils in blood.
- 6. Anemia or thrombocytopenia unresponsive to busulfan/hydroxyurea.
- 7. Persistent thrombocytosis (≥ 1,000,000/ 1) unresponsive to conventional doses of hydroxyurea or busulfan.

- 8. Additional chromosome changes (evolving new clone).
- 9. Increasing splenomegaly unresponsive to conventional doses of hydroxyurea or busulfan.
- 10. Development of chloromas or myelofibrosis.
- 11. Patients in a second (or subsequent) chronic phase after blast crisis.

#### Blastic Phase

1. > 30% blasts plus promyelocytes in the blood or bone marrow.

#### 5.0 **ELIGIBILITY CRITERIA**

#### 5.1 Inclusion Criteria

- 5.1.1 Patients with acute myelogenous or lymphocytic leukemia who are not in first remission or second remission i.e. after failing remission induction therapy or in relapse or beyond second remission, or patients with chronic myelogenous leukemia in blastic phase of the disease are eligible for the study. Patients with refractory anemia with excess blasts and in transformation will be eligible.
- 5.1.2 All candidates for this study must have a HLA (A,B,C,DR) identical siblings who is willing to donate bone marrow for marrow grafting. All ABO blood group combinations of the donor/recipient are acceptable since even major ABO compatibilities can be dealt with by various techniques. (Red cell exchange or plasma exchange). Peripheral blood stem cells or bone marrow can be used.
- 5.1.3 Prior therapy with VP-16 and busulfan is allowed.
- 5.1.4 Patients must be older than 16 and the upper age limit is physiological age of 50.
- 5.1.5 A cardiac evaluation with electrocardiogram and MUGA or echocardiogram is required in all patients. Patients must have an ejection fracture of greater than or equal to 50%.
- 5.1.6 Patients must have a serum creatinine of less than or equal to 1.2 or creatinine clearance > 80ml/min.
- 5.1.7 A bilirubin of less than or equal to 1.5. Patients should also have an SGOT and SGPT less than 5 times the upper limit of normal.
- 5.1.8 Pulmonary function tests including DLCO will be performed. FEV<sub>1</sub> and DLCO should be greater than 50% of predicted normal value.

- 5.1.9 The time from the last induction or reinduction attempt should be greater than or equal to 28 days.
- 5.1.10 Signed informed consent form approved by the IRB is required. The patient, family member and transplant staff physician (physician, nurse, and social worker) meet at least once prior to starting the transplant procedure. During this meeting all pertinent information with respect to risks and benefits to donor and recipient will be presented. Alternative treatment modalities will be discussed. The risks are explained in detail on the enclosed consent forms.

Revised 8/28/00 Revised 3/11/02

Revised 6/13/02

5.1.11 Patients with AML in first remission with poor risk cytogenetics (11q abnormalities, -7,-5, complex abnormalities i.e. > 3 abnormalities, 6;9 translocation and 3q abnormalities del (7q), del (5q), complex abn > abnormalities, 9q, 20q, 21q, 17p, t(9;21).

#### 5.2 Exclusion Criteria

- 5.2.1 Prior radiation therapy that will exclude the use of total body irradiation.
- 5.2.2 Patients who have undergone bone marrow transplantation previously and who have relapsed.
- 5.2.3 Patients with psychological or medical condition that patients physician deems unacceptable to proceed to allogeneic bone marrow transplant.

Revised 8/28/00

5.2.4 Pregnancy

#### 5.3 Donors

- 5.3.1 Any sibling donors who are histocompatible with the prospective recipient will be considered as a suitable donor.
- 5.3.2 Donors will be excluded if for psychological or medical reasons they are unable to tolerate the procedure.
- 5.3.3 Donor should be able to donate peripheral blood stem cells or bone marrow.

#### 6.0 TREATMENT PLAN

All patients will have a right atrial catheter, hickman type inserted. This catheter will be used for collection of blood specimens, administration of drug, bone marrow, blood components, and for hyperalimentation.

- Revised 8/28/00 6.1 Pre-transplant evaluation will be performed within four weeks of beginning treatment except for the following: 1) Bone marrow aspirate and biopsy + cytogenetics within 14 days of starting treatment, 2). CBC, differential, platelets, comprehensive metabolic panel within 5 days of starting treatment.
  - a). Prior to admission patient will have a complete history and physical examination performed. Special attention will be given to prior

chemotherapy, height, weight and body surface area should also be noted.

- b). Patients will have the following laboratory tests performed:
  - CBC with diff platelets i.
  - Sodium, potassium, chloride, bicarbonate or total carbone ii. dioxide, BUN, creatinine, Ca, Mg, Phosphorous, total bilirubin, protein, albumin, SGPT, SGOT. LDH. alkaline phosphatase, cholesterol, glucose.
  - Urine analysis iii.

HIV test

Hepatitis A,B + C

24-hr urine for creatinine clearance

CMV, HSV – HZV ab

Immunoglobulin levels

- İ۷. 24-hour urine collection for creatinine clearance.
- Chest x-ray and EKG ٧.
- CT scan chest, abdomen and pelvis. νi.

Revised 8/28/00

Revised 8/28/00

Rev. 11/8/01

- Pregnancy test vii.
- c). Initial coagulation studies prothrombin time, APTT.
- MUGA scan or echocardiogram d).
- Pulmonary function tests e).
- f). A bone marrow aspirate and biopsy, and cytogenetics needs to be done within 2 weeks of admission (if bone marrow not aspirable and > 20% blasts in blood this may be done on peripheral blood sample).

Patients with acute leukemia or chronic myelogenous leukemia in g).

blast crisis will have a lumbar puncture performed. Methotrexate (10mg/m<sup>2</sup> but not more than a total dose of 12mg) will be administered intrathecally. The spinal fluid will be examined for the presence of malignant cells. Those patients who had leukemic CNS involvement prior to the time of admission before transplantation will receive five weekly intrathecal methotrexate injections with the dose described above from the time patients platelet count is greater than

75,000 to day 100, then monthly intrathecal methotrexate injections with the dose described above between day 100 and 12 months after The initial spinal tap will only be performed if transplantation.

patients platelet count can be kept above 75,000.

#### 6.2 Preparative Chemotherapy Regimen

Rev. 8/12/02

\* Patient to sign consent form before starting Dilantin.

Friday/Day -18

Rev. 11/8/01

Tuesday/Day -14

Begin dilantin 300mg/p.o. t.i.d. times 1 day, then 300mg/p.o./IV daily times 14 days.

Admission or outpatient, dilantin blood levels will be checked and dose adjusted as needed to meet Further adjustments if clinically therapeutic range. indicated. Busulfan test dose administered at 6 a.m. as a single dose. The I/V dose is calculated as follows:

1. Body surface area (BSA) is calculated by the equation:

| BSA=/(Ad | etual body wt.(kg) x height (cm) |
|----------|----------------------------------|
| \/ _ | 3600 |

Rev. 6/13/02

2. 22mg/m<sup>2</sup> I/V Busulfan will be given over 2 hours. Blood levels will be obtained with the first dose as per appendix 1 and will be performed at City of Hope.

Rev. 11/8/01

Wednesday/Day -13

Busulfan AUC will be calculated by standard methods available in the City of Hope Analytical Pharmacology Core Facility (APCF). The resulting AUC will be used to determine the dose required to achieve an AUC of 800 µM\* min according to the following formula:

Adj dose = Current dose x
$$\frac{800\mu\text{Mx min}}{\text{test dose AUC}}$$

Rev. 6/13/02

The maximum dose given will not exceed 32mg/m<sup>2</sup>. There is no limit on dose reduction Busulfan dose will only be adjusted for AUC's <700 or >900 µM\*min.

Thursday/Day -12

The adjusted dose Busulfan dose will be given at 6 a.m. and blood levels will be repeated. Further dose adjustments will be performed if AUC >1000.

Friday/Day -11

Patient admitted to BMT or receive further dose of Busulfan in clinic.

Busulfan dosing restarted at 6 p.m. and is repeated every 6 hours for a total of 14 doses.

Tuesday/Day -7

Fractionated TBI will be given at 120 cGy per fraction for a total of 4 days for a total of 10 fractions for a total dose of 1200 cGy. See Appendix II.

Saturday/Day -3

VP-16 30mg/kg based on adjusted ideal body weight will be administered.

Tuesday/Day 0 PS0

PSC reinfusion/or BM infusion

See Appendix 3 for PSC Collection

Toxicities of the marrow infusion are very rare. Volume overload may be prevented by removal of plasma from the marrow aspirate or by phlebotomy of the recipient prior to marrow infusion. Pulmonary emboli are theoretically possible and would require management with 02 or IPPB. However, our clinical observations over the last 20 years indicate that pulmonary embolism in this clinical setting does

not occur at any increased rate. The most frequently encountered problem is that of chills, hives, and fever. Those allergic reactions occur rarely (in 1 to 2%) and can be prevented by intravenous injections of dyphenhydrimine 25mg and hydrocortisone (50mg) prior to the bone marrow infusion.

#### 6.3 Recommended

6.3 Graft Versus Host Disease Prophylaxis and Treatment

#### MMF

Both intravenous and oral doses of MMF will be calculated using adjusted ideal body weight. If actual body weight is less than ideal body weight, actual body weight will be used. All patients will initiate the intravenous formulation of MMF on the day of transplantation (Day 0), a minimum of 2 hours after the end of the stem cell infusion. MMF will be administered at 30mg/kg/day in two divided daily doses from day 0 until day 27. At day 27 the MMF will be tapered by 250mg to be off by Day 56. If patient does not develop evidence of GVH. The intravenous formulation will be administered until at least day 14 after transplant. MMF will be administered as a 2 hour IV infusion. MMF will be induced with 5% dextrose. When patients have recovered from radiation-induced gastroenteritis and are capable of taking the oral MMF, they will be converted at an oral to intravenous ratio of 1:1. This can be done because of the high bioavailability of MMF. The oral formulation of MMF is available in 250mg capsules. The prescribed dose will be rounded to the nearest dose possible with these capsules.

Revised 6/13/02

#### 2. Cyclosporine

All patients will receive cyclosporine 3mg/kg/day IV or 12.5 mg/kg/day orally from day –1 until day 50. Dosing should be based on adjusted ideal body weight. If GVHD is absent, cyclosporine will then be tapered by 5% week until day 180 when the drug is discontinued. Cyclosporine whole blood levels will be monitored.

- 6.31 If moderate to severe graft-versus-host disease occurs (Grade II-IV), patients will be treated with the administration of higher doses of methylprednisolone, anti-thymocyte globulin, etc.
- 6.32 Graft-versus-host disease will be graded according to previously defined criteria (Appendix IV,V).

#### 6.4 Supportive Care during Transplant

On the day of admission menstruating females will start Provera 10mg p.o. daily and Nystatin vaginal suppositories 1 b.i.d. In addition, all patients will start, levofloxacin 500mg/p.o or I/V q daily, Bactrim DS 1 tablet p.o. b.i.d. or IV will be started and continue until day –2.

Hyperalimentation will be given while patient is unable to eat.

It is recommended that platelet transfusions will be given to maintain platelet count greater than 20,000/µl at all times. Single donor platelets will be used with an attempt to use family members when possible. All platelets will be filtered to remove contaminated leukocytes which may harbor cytomegalovirus (CMV). Packed RBC transfusions will be used to keep the hemoglobin greater than 8.5gm/dl. All blood products will be irradiated with 2500cGy prior to tranfusions.

The management of infections in these immunocompromised patients must by necessity be individualized, but the following general approach will be utilized. If a specific infection is documented, patients will be placed on specific anti-microbial agents to treat that infection. For temperatures greater than 38.5°C without an obvious source in patients with less than 1000granulocytes/I, cultures of blood will be obtained. Following this, a third generation cephalosporin will be used as initial empiric antibiotic coverage. For persistent or recurrent fevers an aminoglycoside and or ancef will be added. Prophylactic intravenous amphotericin B will be used and the dose can be increased as clinically indicated. If a specific organism or site of infection is identified after starting empiric antibiotic coverage, therapy will be changed as needed.

Rev. 11/8/01

While hospitalized, patients will have daily CBC's with platelet count, and SMA-7 (Na, K, C1, CO<sub>2</sub>, BUN, creatinine, glucose). SMA12 (total protein, albumin, phosphatase, Ca, SGPT, SGOT, alkaline phosphatase, total bilirubin, cholesterol) determinations will be performed on Monday, Wednesday and Fridays and chest x-rays will be done weekly. CSA levels q Mon & Thurs, and CMV blood cultures q Mon & Thurs when WBC >2000.

#### 7.0 TOXICITIES TO BE MONITORED AND DOSAGE MODIFICATIONS

- 7.1 Radiation toxicities: The short term complications of TBI are: a). nausea and vomiting. This problem will be managed symptomatically. b) Oral mucositis is expected in all patients. All patients will receive oral care with hydrogen peroxide and clotrimazole. Only sponge toothbrushes will be allowed. Pain will be managed with morphine and dilaudid, c) Temporary alopecia will also be expected in all patients. Long-term complications of TBI include: a) cataracts, these can be managed successfully in the same way as cataracts unrelated to radiation. b) Solid tumors have been seen following TBI. c) Radiation fibrosis of the lungs, d) hypothyroidism and patient will be required to take supplemental thyroid medication, e). Sterility.
- 7.2 Chemotherapy Toxicities:
  - 7.2.1 Toxicities of VP-16
    - a) VP-16 may cause nausea, vomiting lasting for a few hours.
    - b). Occassionally VP16 can cause allergic reactions, hemorrhagic cystitis and hepatotoxicity.
    - b) Can cause mucositis, and dermatitis.
  - 7.2.2 Busulfan Toxicities are myelosuppression, pulmonary fibrosis, increased pigmentation, grand mal seizures and temporary or permanent alopecias have also been seen.

If 2 of first 6 patients develop grade 3 liver or lung toxicity related to the preparative regimen the Busulfan dose will be decreased to the equivalent of 9mg/kg of the oral dose and AUC range will be changed to 600-800.

If 2 of first 6 patients require ventilator support for mucositis the VP-16 will be omitted.

7.3 The dose of methotrexate will be modified for impaired liver function based on serum direct bilirubin as follows:

| Direct Bilirubin mg/dl | % MTX dose |
|------------------------|------------|
| ₹2 | 100% |
| 2.1 - 3.0 | 50% |
| > 3.0 | 0% |

7.4 The dose of cyclosporine and methotrexate will be modified for impaired renal function based on serum creatinine.

| Creatinine mg/dl | % CSA + MTX |
|------------------|-------------|
| < 1.5 | 100% |
| 1.6 – 1.7 | 75% |
| 1.8 - 2.0 | 50% |
| > 2.0 | 0% |

- Toxicities will be graded per CTC 2.0 (Appendix VII) publish date April 30, 1999.  $^{
  m Rev.~11/8/01}$ 0.8
- 9.0 STUDY CALENDAR SEE APPENDIX VI.

#### CRITERIA FOR EVALUATION AND DEFINITION

- 10.1 Achievement of a lymphohematopoietic graft is defined as recovery from posttransplant.
- 10.2 Complete remission is defined as attainment of M-1 marrow status, and no evidence of recurrent extramedullary disease.
- 10.3 Length of survival is measured from entry on study to death or time of last contact.
- Treatment failure is defined as death from toxicities associated with transplant 10.4 procedure of recurrence of malignancy.
- 10.5 All registered patients including those removed from the treatment protocol will be followed for survival every six months.

#### 11.0 CRITERIA FOR REMOVAL FROM STUDY

There are two situations that will determine removal of a patient from the study:

- 11A. The patient may always be removed from the study whenever he/she wishes.
- 11B. If the scheduled bone marrow donor decides not to provide bone marrow.

#### 12.0 STATISTICAL CONSIDERATIONS

12.1 Primary and Secondary Endpoints: The primary endpoint of the Phase II study is to evaluate the efficacy of FTBI/BU/VP-16 with a targeted Busulfan dose of AUC 700-900 as a preparative regimen for allogeneic BMT in patients with advanced hematological malignancies (AML or ALL beyond second remission, in induction failure, or in relapse; CML in blast crisis; and myelodysplasia, RAEB and RAEBIT). Secondary endpoints will include early and late toxicities of this regimen.

Efficacy will be estimated based on 2 and 5 year disease-free survival (DFS). The effects of cytogenetics, WBC at presentation, and number of courses of induction therapy to achieve remission will be evaluated as possible prognostic factors for relapse, DFS, and overall survival.

- 12.2 <u>Sample size Estimation and Length of Accrual</u>: A total of 50 patients with advanced malignancies and less than 50 years old (physiological age) will be accrued to this trial, so that in estimating the engraftment and relapse rates the maximum standard error will be 0.7. We expect to accrue approximately 10-12 patients per year so that this trial will require 4-5 years of completion.
- 12.3 If at any time the severe treatment related complication rate (e.g. severe VOD, interstitial pneumonia, neurotoxicity at day 100 post BMT) or regimen related mortality exceeds 20% with a high probability (i.e. >95%) then further accrual to the trial will be terminated. This would occur if the following numbers of events have been observed, monitoring after every set of 10 patients is accrued:

| Number of Patients | Number of Events Leading to Early |
|--------------------|-----------------------------------|
| Accrued | Termination |
| 10 | 5 |
| 20 | 8 |
| 30 | 11 |
| 40 | 14 |

12.4 <u>Statistical Analyses</u>: The rate of engraftment and median time to engraftment will be estimated, defined as time to ANC > 500 and platelets >20,000.

The Kaplan-Meier method will be used to estimate time to relapse, DFS, and overall survival, and 95% confidence intervals will be calculated using Greenwood's variance.

The intent-to-treat group will include all patients receiving the preparative regimen for BMT. For overall survival, failure time will be calculated from the day of first treatment to the day of death due to any cause for those patients who fail. For DFS, the failure time will be calculated from the day of first treatment to the day of disease relapse or death due to any cause. For patients who remain alive and well at the time of analysis, the survival time will be censored as of the date of last contact. The Cox proportional hazard regression model will be used to analyze possible prognostic factors for relapse, DFS and overall survival.

Revised 9/26/00

12.5 Patients with AML with unfavorable cytogenetics will be a subset analysis that will include approximately 12 patients. This number is too small for formal hypothesis testing. It will give us some experience with this population of patients and descriptive analysis will be used along with estimation of relapse rate and 95% C.I.

#### 13.0 WOMEN AND MINORITIES GUIDELINES

All eligible patients from both genders and from all racial/ethnic groups will be recruited equally into this trial, with the only exclusionary criteria being those stated in Section 5.0. Based on our patient populations and previous experience with BMT for advanced hematological malignancies, the anticipated rates of entry into this study by gender and race/ethnicity are as follows:

## Race/Ethnicity by Gender for Advanced Malignancy Patients Receiving BMT at City of Hope

| | American<br>Indian or<br>Alaskan<br>Native | Asian or<br>Pacific<br>Islander | Black, not of<br>Hispanic<br>Origin | Hispanic | White, not<br>of Hispanic<br>Origin | Other or unknown |
|---|---|---|---|---|---|---|
| Female | 0% | 8% | 1% | 32% | 58% | 1% |
| Male | <1% | 8% | 3% | 33% | 54% | 3% |
| Total | <1% | 8% | 2% | 33% | 55% | 2% |

99041 - Version 07 4/20/04

14.0 <u>GUIDELINES FOR REPORTING ADVERSE EVENTS (AE) ADVERSE DRUG REACTIONS ADR OCCURRING WITH COMMERCIAL AGENTS. APPENDIX VIII.</u>

Rev. 11/8/01

#### 15.0 REFERENCES:

- 1. Slattery JT, Clift RA, Buckner CD, et al. Marrow transplantation for chronic myeloid leukemia: The influence of plasma busulfan levels on the outcome of transplantation. Blood 1997; 89:3055-3060.
- 2. Snyder DS, Negrin RS, O'Donnell MR, et al. Fractionated total body irradiation and high dose etoposide as a preparatory regimen for bone marrow transplantation for 94 patients with chronic myelogenous leukemia. Blood 1994;84: 1672-1679.
- 3. Clift RA, Buckner CD, Thomas ED, et al. Marrow transplantation for chronic myeloid leukemia: A randomized study comparing cyclophosphamide and total body irradiation with busulfan and cyclophosphamide. Blood 1994; 84: 2036-2043.
- 4. McGlave PB, Haake RJ, Bostrom BC, et al. Allogeneic bone marrow transplantation for acute nonlymphocytic leukemia in first remission. Blood 1988;72: 1512-1517.
- 5. Forman SJ, Spruce WE, Farbstein MJ, et al. Bone marrow ablation followed by allogeneic marrow grafting during first complete remission of acute nonlymphocytic leukemia. Blood 1983; 61:439-442.
- 6. Blume KG, Beutler E, Bross KJ, et al. Bone-marrow ablation and allogeneic marrow transplantation in acute leukemia. N Engl J Med 1980;302:1041-1046.
- 7. Blume KG, Forman SJ, Krance RA, Henke M, Findley DO, Hill LR. Bone marrow transplantation for acute leukemia. Hematol Blood Transfusion 1985; 29:39-41.
- 8. Thomas ED, Sanders JE, Flournoy N, et al. Marrow transplantation for patients with acute lymphoblastic leukemia in remission. Blood 1979;54:468-476.
- 9. Martin PJ, Clift RA, Fisher LD, et al. HLA-identical marrow transplantation during accelerated phase chronic myelogenous leukemia: Analysis of survival and remission duration. Blood 1988;72:1978-1984.
- 10. Clift RA, Buckner CD, Thomas ED, et al. Marrow transplantation for patients in accelerated phase of chronic myeloid leukemia. Blood 1994;84:4368-4373.
- 11. Mehta J, Powles R, Horton C, et al. Bone marrow transplantation for primary refractory acute leukemia. Bone Marrow Transplant 1994;14:415-418.
- 12. Forman SJ, Schmidt GM, Nademanee AP, et al. Allogeneic bone marrow transplantation as therapy for primary induction failure for patients with acute leukemia. J. Clin Oncol 1991;9:1570-1574.
- 13. Clift RA, Buckner CD, Appelbaum FR, et al. Allogeneic marrow transplantation during untreated first relapse of acute myeloid leukemia. J. Clin Oncol 1992;10:1723-1729.
- 14. Appelbaum FR, Clift RA, Buckner CD, et al. Allogeneic marrow transplantation for acute nonlymphoblastic leukemia after first relapse. Blood 1983;61:949-953.

- 15. Blume KG, Forman SJ, O'Donnell MR, et al. Total body irradiation and high-dose etoposide: A new preparatory regimen for bone marrow transplantation in patients with advanced hematologic malignancies. Blood 1987;69:1015-1020.
- 16. Tutschka PJ, Copelan EA, Klein JP. Bone marrow transplantation for leukemia following a new busulfan and cyclophosphamide regimen. Blood 1987;70: 1382-1388.
- 17. Clift RA, Buckner CD, Appelbaum FR, et al. Allogeneic marrow transplantation in patients with acute myeloid leukemia in first remission: A randomized trial of two irradiation regimens. Blood 1990;76: 1867-1871.
- 18. Santos GW, Tutschka PJ, Brookmeyer R, et al. Marrow transplantation for acute nonlymphocytic leukemia after treatment with busulfan and cyclosphosphamide. N Engl J Med 1983;309:1347-1353.
- 19. Brown RA, Wolff SN, Fay JW, et al. High-dose etoposide, cyclophosphamide, and total body irradiation with allogeneic bone marrow transplantation for patients with acute myeloid leukemia in untreated first relapse: A study by the North American Marrow Transplant Group. Blood 1995;85:1391-1395.
- 20. Demirer T, Buckner CD, Appelbaum FR, et al. Busulfan, cyclophosphamide and fractionated total body irradiation for allogeneic marrow transplantation in advanced acute and chronic myelogenous leukemia: Phase I dose escalation of busulfan based on targeted plasma levels. Bone Marrow Transplant 1996;17:341-346.
- 21. Snyder DS, Chao NJ, Amylon MD, et al. Fractionated total body irradiation and high-dose etoposide as a preparatory regimen for bone marrow transplantation for 99 patients with acute leukemia in first complete remission. Blood 1993;82:2920-2928.
- 22. Blume KG, Kopecky KJ, Henslee-Downey JP, et al. A prospective randomized comparison of total body irradiation-etoposide versus busulfan-cyclophosphamide as preparatory regimens for bone marrow transplantation in patients with leukemia who were not in first remission: A Southwest Oncology Group study. Blood 1993; 81:2187-2193.
- 23. Linker CA, Ries CA, Damon LE, Rugo HS, Wolff JL. Autologous bone marrow transplantation for acute myeloid leukemia using busulfan plus etoposide as a preparative regimen. Blood 1993; 81: 311-318.
- 24. Chao NJ, Stein AS, Long GD et al. Busulfan/Etoposide-Initial experience with a new preparatory regimen for autologous bone marrow transplantation in patients with acute non-lymphoblastic leukemia. Blood 1993; 81: 319-323.
- 25. Kashyap, S.J. Forman, P. Cagnoni, H. Fernandez, W. Hu, V. Gian, J. Wingard, S. Tarantolo, B.S. Andersson. (1998) Intravenous Busulfan (Busulfex™)/Cytoxan (CY) Preparative Regimen for Allogeneic (ALLO) and Autologous (AUTO) Hematopoietic Stem Cell Transplantation (BMT) is well Tolerated by Patients Over 50 Years of Age. ASH, December 1998, Miami Beach
- 26. W.P. Vaughan, P. Cagnoni, H. Fernandez, W. Hu, A. Kashyap, V. Gian\*, J. Wingard, S. Tarantolo, B.S. Andersson (1998) Decreased Incidence of and Risk Factors for Hepatic

Veno-Occlusive Disease with an Intravenous Busulfan (BU) Containing Preparative Regimen for Hematopoietic Stem Cell Transplantation (HSCT). ASH, December 1998, Miami Beach

- 27. B.S. Andersson, K. McWilliams, H. Tran, H. Fernandez, P. Cagnoni, R. Jones, V. Gian, S. Tarantolo, A. Kashyap, S.J. Forman, WW Hu, KG Blume, R.E. Champlin (1998) IV Busulfan, Cyclosphosphamide (Bu/Cy) and Allogeneic Hemopoietic Stem Cells (BMT) for Chronic Myeloid Leukemia (CML), ASH, December 1998, Miami Beach
- Vaughan WP, Soong S, Cagnoni P, Fernandez H, et al. Body surface area (BSA) Dosing using actual body weight (ABW) yields less variation in Area under the concentration x time curve (AUC) for high dose I/V Busulfan (Bu) than BSA dosing using ideal body weight (IBW), Adjusted ideal body weight (AIBW) or dosing using ABW, IBW or AIBW directly.

  ASCO, May 15- 19, 1999

# APPENDIX I IV BUSULFAN KINETICS FORM

| IRB#: | DATE: | (CIRCLE WEIGHT USED) |
|---------------------|-------------|----------------------|
| PATIENT | DOSE # | Actual Body Weight |
| Medical Record # | Start time: | Ideal Body Weight |
| MD/Pager # | Stop Time: | Adjusted IBW |
| Coordinator/Pager # | DOSE:mg | |

#### INFUSION TO RUN OVER 2 HOURS

| Tube # | Collection Schedule | Proposed Collection Time Actual Collection Time |
|---|---|---|
| 1 | Immediately prior to beginning of infusion | APPROX. 0555 |
| 2 | Immediately prior to end of infusion | APPROX. 0755 |
| 3 | 15 minutes post infusion | APPROX. 0815 |
| 4 | 30 minutes post infusion | APPROX. 0830 |
| 5 | 60 minutes post infusion (1 hour) | APPROX. 0900 |
| 6 | 180 minutes post infusion (3 hours) | APPROX. 1100 |
| 7 | 240 minutes post infusion (4 hours) | APPROX. 1200 |

<sup>\*\*</sup> ALL samples to be obtained in 7cc green top tubes (Sodium Heparin) and kept on ice at Nurses Station.

| Then send to Clinic | cal Pathology. |
|---------------------|----------------|
| RN SIGNATURE _ | |

Appendix II

#### FRACTIONATED TOTAL BODY IRRADIATION SCHEMA

| Session | Day | Time | Beam<br>Direction | Energy (MeV) | Dose (rads) | Notes |
|---|---|---|---|---|---|---|
| 1 | -7 | 0730 | AP | 8/10X | 120 | TLD |
| | | | AP | Electron | | Testes male |
| | | | | | | (ALL only) |
| 2 | -7 | 1200 | AP | Electron | 400 | TLD |
| 3 | -7 | 1630 | PA | 8/10X | 120 | |
| 4 | -6 | 0730 | AP | 8/10X | 120+ | (PA Chestwall |
| | | | | | | Boost) 300 |
| 5 | -6 | 1200 | PA | 8/10X | 120+ | (AP Chestwall |
| | | | | | | Boost) 300 |
| 6 | -6 | 1630 | AP | 8/10X | 120 | · |
| 7 | -5 | 0730 | AP | 8/10X | 120 | |
| | | | AP | electron | 300 | Chest wall boost |
| 8 | -5 | 1200 | PA | 8/10X | 120+ | (PA Chestwall |
| | | | | | | Boost -300) |
| 9 | -5 | 1630 | PA | 8/10X | 120 | , |
| 10 | -4 | 0730 | PA | 8/10X | 120 | |

Photon dose is calculated at mid-depth, central axis. Electron chest wall dose is calculated at 90% isodose level, where electron energy is selected to place 90% isodose level at pleural surface. At the first AP and PA sessions for total body irradiation, portal films with the treatment beam will be obtained prior to treatment to assure proper lung block placement. The x-ray total body irradiation dose given during portal film will be subtracted from the total dose planned for that session. Subsequent placement of lung blocks at the remaining sessions will be documented by verification films obtained during the actual treatment.

During the first AP and PA sessions for total body irradiation, the radiation dose received by the patient will be monitored by means of thermoluminescent dosimeters placed on the anterior surface of the patient's skin at the following anatomic locations: forehead, suprasternal notch, xiphoid process, umbilicus, pelvis, mid-thigh, knee, mid-calf, and ankle. The midline dose to the patient can be calculated from the sum of entrance and exit doses recorded by the thermoluminescent dosimeter. If thermoluminescent dosimeter indicates a deviation of greater than  $\pm$  10% in the planned dose, either the compensating filter, the machine monitor units, or both may be modified for subsequent sessions.

#### Appendix III

- 1). G-CSF Administration to Donors: All donors will receive G-CSF 10 μg/kg/day for 6 consecutive days from day –5 to day 0. G-CSF will be administered by a subcutaneous injection daily beginning 5 days prior to day 0 (defined as the day marrow would ordinarily be given).
- 2). <u>PBSC Collection</u>: Donors may undergo vein to vein collections or may receive an appropriate catheter inserted on or before day of the treatment regimen. Donors will receive -5 daily doses of G-CSF, 10µg/kg/day by subcutaneous injection commencing on day -5. These doses will be administered each day in the Outpatient Department or at home.

Treatment Schema for Donor

| Days | -5 | -4 | -3 | -2 | -1 | 0 |
|------------------|----|----|----|----|----|---|
| G-CSF 10µg/kg/SQ | Х | Χ | Χ | Χ | Х | |
| PBSC Collection | | | | | Х | Χ |

PBSC's will be collected in the afternoon of day -1 and reinfused on day 0. \*If the collection on day -1 contains less than  $5.0 \times 10^6$  CD34+ cells per kg recipient weight, a second collection will be performed the following morning and transfused on day 0.

If PBSC's cannot be collected by a vein to vein technique, a percutaneous Mahurkar catheter will be inserted.

General procedures will include the use of a standard apheresis machined (COBE Spectra, Lakewood Colo.), and processing up to 16 I of whole blood during the collection. (Refer to Standard Practice Manual for collection procedure).

### APPENDIX IV

#### Acute Graft Versus Host Disease Staging and Grading Table

### Clinical Stage of acute GVHD according to Organ System

| Stage | Skin | Liver | Intestine |
|---|---|---|---|
| + | Maculopapular rash <25% of | Bilirubin 2-3mg/dl | >500-1000 ml diarrhea per |
| | body surface | | day or (nausea, anorexia or |
| | | | vomiting with biopsy (EGD) |
| | | | confirmation of upper GI |
| | | | GVHD |
| ++ | Maculopapular rash 25-50% | Bilirubin 3-6mg/dl | >1000-1500 ml diarrhea per |
| | of body surface | | day |
| +++ | Maculopapular rash >50% | Bilirubin 6-15mg/dl | >1500 ml diarrhea per day |
| | body surface area or | | |
| | Generalized erythroderma | | |
| ++++ | Generalized erythroderma | Bilirubin >15mg/dl | >1500 ml diarrhea per day |
| | with bullous formation and | _ | plus severe abdominal pain |
| | desquamation | | with or without ileus |

### Overall Clinical Grading of Severity of acute GVHD

| Grade | Skin | Liver | GI |
|-----------------------------|------|------------------|-----|
| I | 1-2 | 0 | 0 |
| $\mathrm{II}^{\mathrm{A}}$ | 0 | 0-1 | 1 |
| | 0 | 1 | 0-1 |
| | 1-3 | 0-1 | 1 |
| | 1-3 | 1 | 0-1 |
| | 3 | 0 | 0 |
| $\mathrm{III}^{\mathrm{A}}$ | 0-3 | 2-3 | 0-2 |
| | 0-3 | 0-3 | 2-3 |
| | 0-3 | $4^{\mathrm{B}}$ | 0-3 |
| $IV^{A}$ | 0-3 | 0-4 | 4 |
| | 4 | 0-4 | 0-4 |

- A. Grade II-IV GVHD with only single organ involvement should be biopsy confirmed.
- B. If Karnofsky performance status is  $\leq 30\%$ , then Grade IV.

#### APPENDIX V

#### Grading of Chronic Graft Versus Host Disease

Definitions:

<u>Progressive</u>: Direct continuation from preceding acute GVHD.

Quiescent: Arising after complete resolution of acute GVHD.

de Novo: No preceding GVHD.

Subclinical disease: Characteristic pathology findings on both blind oral and skin biopsies in

absence of clinical signs or symptoms.

<u>Clinical disease:</u> Multi-organ clinical manifestations and positive skin and oral biopsies

<u>Limited cGVHD</u>: Either or both of the following:

1. Localized skin involvement

2. Hepatic dysfunction due to cGVHD

Extensive cGVHD: Either

1. Generalized skin involvement

2. Localized skin involvement and/or hepatic dysfunction due to chronic GVHD

#### **PLUS**

- 3. Liver histology showing chronic aggressive hepatitis, bridging necrosis or cirrhosis, OR
- 4. Eye involvement with Schirmer's test with less than 5 mm wetting, OR
- 5. Positive lip biopsy
- 6. Involvement of any other target organ

Reference: Chronic Graft Versus Host Disease: Pathology, diagnosis, treatment and prognostic

factors, BMT – Exp Hem Today 1988

#### APPENDIX VI

| Studies adm -17 -13 -12 -11 -10 -9 -8 -7 -6 -5 -4 -3 -2 -1 0 1 2 3 4 6 7 100 180 | HD Therapy/ | Fransp | | | | | | ept BM | | | | | | | | | | rior to | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| The control of the | Required | Pre | Day | Day | | | Day | Day | Day | Day | Day | Day | Day | Day | Day | Day | Day | Day | Day | Day | Day | Day | Day | Day | Day | Yearly |
| CBC.DHIF, PI.T=+++ | studies | adm | -17 | -13 | -12 | -11 | -10 | -9 | -8 | -7 | -6 | -5 | -4 | -3 | -2 | -1 | 0 | 1 | 2 | 3 | 4 | 6 | 7 | 100 | 180 | X 2 |
| PIT-++ | | | | | | | | | | | | | | | | | | | | | | | | | | years |
| Sma-1 | | X | X | X | X | X | X | | | | X | | | | X | | X | X | X | X | X | | | X | | X |
| SMA-12 ++ | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Hepatitis a,b,c | | | | X | | X | | | | | X | | | | | | X | | X | | X | | | | | X |
| Hepatitis a,b,c X | | | | | | | | | | | | | | | | | | X | | X | | | | X | | X |
| HIV | | | X | | X | | X | | | | | | | | X | | | | X | | | | | | | |
| PT.PTT | | | | | | | | | | | | | | | | | | | | | | | | | | |
| UA | | | | | | | | | | | | | | | | | | | | | | | | | | |
| 24hr Crea cl X | PT,PTT | X | | | | | | | | | | | | | | | | | | | | | | | | |
| Pregnancy test | UA | X | | | | | | | | | | | | | | | | | | | | | | | | |
| CMV,HSV/HZ | 24hr Crea cl | X | | | | | | | | | | | | | | | | | | | | | | | | |
| CMV,HSV/HZ | Pregnancy test | X | | | | | | | | | | | | | | | | | | | | | | | | |
| Immunoglobulin X | | | | | | | | | | | | | | | | | | | | | | | | | | |
| PFT | | | | | | | | | | | | | | | | | | | | | | | | | | |
| PFT | Immunoglobulin | X | | | | | | | | | | | | | | | | | | | | | | | | |
| ++CXR X | _ | | | | | | | | | | | | | | | | | | | | | | | | | · |
| ++CXR X | EKG | X | | | | | | | | | | | | | | | | | | | | | | | | |
| CT Scan Chest, ABD | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Chest, ABD Che | | | | | | | | | | | | | | | | | | | | | | | | | | |
| ECHO or MUGA | | 11 | | | | | | | | | | | | | | | | | | | | | | | | |
| MUGA | | X | | | | | | | | | | | | | | | | | | | | | | | | |
| LP see 6.1g X | | 11 | | | | | | | | | | | | | | | | | | | | | | | | |
| BM asp, bx, cytogenetics | | X | | | | | | | | | | | | | | | | | | | | | | | | |
| Dilantin level | | | | | | | | | | | | | | | | | | | | | | | | X | | X |
| Dilantin level | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Busulfan levels | | | | X | | | | | | | | | | | | | | | | | | | | | | |
| TREATMENT Image: Control of the control o | | | | | | XX* | | | | | | | | | | | | | | | | | | | | |
| Dilantin X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X< | 240411411101010 | | | 2121 | | * | | | | | | | | | | | | | | | | | | | | |
| Dilantin X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X< | TREATMENT | | | | | | | | | | | | | | | | | | | | | | | | | |
| Busulfan X X** X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X | | T <sup>'</sup> | X | X | X | X | X | X | X | X | X | X | X | | | | | | | | | | | | | |
| FTBI X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X | | | | | | | | | | | | | | | | | | | | | | | | | | |
| VP-16 X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X <td></td> <td></td> <td></td> <td></td> <td><del></del></td> <td></td> <td></td> <td>1</td> <td></td> <td></td> <td>X</td> <td>X</td> <td>X</td> <td>x</td> <td></td> <td></td> <td></td> <td></td> <td></td> <td>t</td> <td></td> <td></td> <td></td> <td>t</td> <td></td> <td></td> | | | | | <del></del> | | | 1 | | | X | X | X | x | | | | | | t | | | | t | | |
| PSC's or BM X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X <td< td=""><td></td><td></td><td></td><td></td><td>1</td><td></td><td></td><td></td><td></td><td>1</td><td></td><td></td><td></td><td></td><td>x</td><td></td><td></td><td></td><td>1</td><td>1</td><td></td><td></td><td></td><td>1</td><td></td><td></td></td<> | | | | | 1 | | | | | 1 | | | | | x | | | | 1 | 1 | | | | 1 | | |
| CNS Disease | | | | | | | | | | | | | | | 21 | | X | | | | | | | | | |
| | | | | | | | | - | | | | - | - | | - | | 71 | | | - | | | - | - | | |
| patients see | | | | | | | | | | | | | | | | | | | | | | | | | | |
| section 6.53 | section 6.53 | | | | | | | | | | | | | | | | | | | | | | | | | |

<sup>\$</sup> Dilantin will be given daily consecutively until day -14

28 Rev. 11/8/01

<sup>++</sup> Every Monday, Wednesday, Friday during hospitalization, CXR to be done weekly XX blood sample shipment

<sup>\*\*</sup> If required

#### **APPENDIX VII**

CTC Version 2.0 Publish Date: April 30, 1999

## COMMON TOXICITY CRITERIA (CTC)

| | Grade Adverse Event 0 1 | | | |
|---|---|---|---|---|
| 0 | 1 | 2 | 3 | 4 |
| | ALLERGY/IN | MMUNOLOGY | | |
| Done | transient rash, drug<br>fever <38°C (<100.4°F) | urticaria, drug fever 238°C (2100.4°F), and/or asymptomatic broachospasm | symptomatic bronchospa sm. requiring parenteral medication(s), with or without urticaria; allergy-related edema/angioedema | anaphylaxis |
| none | muld, not requiring treatment | moderate, requiring treatment | raded in the DERMATOLO | GY/SKIN category. |
| none | serologic or other evidence of autoimmune reaction but patient is asymptomatic (e.g., viciligo), all organ function is normal and no treatment is required | evidence of autoimmune reaction involving a non-essential organ or function (e.g., bypothyroidism), requiring treatment other than immunosuppressive drugs | reversible autoimmune reaction involving function of a major organ or other adverse event (e.g., transient colitis or anemia), requiring short-term immunosuppressive treatment | autoimmune reaction causing major grade 4 organ dysfunction; progressive and irreversible reaction: long-term administration of high dose immunosuppressive therapy required |
| | lobia. Hemolysis. | | | |
| | * | • | present | - |
| e as Allergic reac | tion/hypersensitivity above. | ited symptom. If it occurs v | with other manifestations of | allergic or |
| DODE | mild, not requiring<br>treatment | symptomatic, requiring medication | requiring steroids | ischemic changes or<br>requiring amputation |
| DODE | mild | moderate | Severe | life-threatening or<br>disabling |
| | AUDITORY | /HEARING | | |
| ed as Middle ear | hearing in the AUDITORY/HEAR | LING category. | | |
| category. | · | | | <del></del> |
| normal | external otitis with<br>erythema or dry<br>desquamation | external oditis with<br>moist desquamation | external oticis with<br>discharge, massoiditis | necrosis of the canal<br>soft tissue or bone |
| | Done absence of other Done Done MATOLOGY/SI e as Allergic read Done Done das Middle ear | ALLERGY/IT Bone transieut rash, drug fever <38°C (<100.4°F) absence of other manifestations of an altergic or by mild, not requiring treatment Bone serologic or other evidence of autoimmune reaction but patient is asymptomatic (e.g., vitiligo), all organ function is normal and no treatment is required Colitis, Hemoglobin, Hemolysis, Bone | ALLERGY/IMMUNOLOGY bone transient rash, drug fever <38°C (<100.4°F) 28°C (≥100.4°F). and/or asymptomatic bronchospasm absence of other manifestations of an allergic or hypersensitivity reaction, is gone mild, not requiring treatment treatment treatment autoimmune reaction involving a non-evidence of autoimmune reaction involving a non-but patient is asymptomatic (e.g., vitilgo), all organ function is normal and no treatment is required other than immunosuppressive drugs Colitis, Hemoglobia, Hemolysis. Bone MATOLOGY/SKIN category if it occurs as an isolated symptom. If it occurs as a Allergic reaction/hypersensitivity above. Bone mild not requiring symptomatic, requiring treatment medication moderate AUDITORY/HEARING ed as Middle ear/hearing in the AUDITORY/HEARING category. Dormal external otitis with external otitis with moist desquarmation | ALLERGY/IMMUNOLOGY Bone transient rash, drug fever <38°C (<100.4°F), and/or symptomatic bronchospasm requiring parenteral medicition(s), with or without urricara; allergy-related edema/angioedema edema/angioedema reaction involving a none serologic or other evidence of autoimmune reaction involving a none bus patient is asymptomatic (e.g., vitiligo), all organ function is normal and no treatment is required and no treatment is required bronchospasm requiring parenteral medicition(s), with or without urricara; allergy-related edema/angioedema evidence of autoimmune reaction involving a non-essential organ or function of a major organ or other adverse organ or other adverse organ or other adverse organ or other adverse organ or other adverse drugs freatment colitis or anemia), requiring treatment colitis or anemia), requiring storit-term immunosuppressive drugs Colitis. Hemoglobia. Hemolysis. Done MATOLOGY/SKIN category if it occurs as an isolated symptom. If it occurs with other manifestations of a sa Allergic reaction/hypersensitivity above. Done mild moderate severe AUDITORY/HEARING external otitis with external otitis with moist desquarmation discharge, massoiditis |

| | | C | rade | | |
|---|---|---|---|---|---|
| Adverse Event | a | 1 | √2 × √ | 3 | 4 |
| laner eur/hearing | oormai .·· | bearing loss on<br>audinmetry only | tinging or bearing loss, not requiring bearing and or treatment | tinulus or bearing loss,<br>correctable with hearing<br>aid or treatment | severe unilateral or bilateral hearing loss (deafess), not correctable |
| Middie ear/bearing | pormal | serous otitis without<br>subjective decrease in<br>hearing | serous otics or infection requiring medical intervention; subjective decrease in hearing; rupture of tympanic membrane with discharge | ocitis with discharge,<br>massoiduis or<br>conductive hearing loss | necrosis of the canal<br>soft tissue or bone |
| Auditory/Hearing - Other (Specify: | pormal | mild | moderate | severe | life-durencening or<br>disabling |
| | _ | BLOOD/BO | NE MARROW | | No. |
| Bone marrow cellularity | normal for age | mildly hypocellular or \$25% reduction from normal cellularity for age | moderately hypocellular or >25 - <50% reduction from normal cellularity for age or >2 but <4 weeks to recovery of normal bone marrow cellularity | severely hypocellular or >50 - \$75% reduction in cellularity for age or 4 - 6 weeks to recovery of normal bone marrow cellularity | aplasia or >6 weeks to recovery of normal bone marrow cellularity |
| Normal ranges: | | | | | |
| children (SI8 years) | 90% rellularity | frig 12 chengering griffen reeren fifterengartige fere eriffengig | | | |
| younger adults (19-59) | 50 - 70%<br>cellularity average | and a supplementable of the effects of the supplementable of the s | المنطق في منصور فا وسائيك من هندس بي كيري و من و و هن من وطائق في فو رسان دفق بنا | ود د عود محمود چه دو د چه و مودو خستر ده مد څه څه کو د موملوگونو و و د شد پر سیمند وټه نیونه | |
| older adults (≥60 years) | 50% cellularity average | | | | |
| Note: Grade Bose marrow cel | llularity only for change | s related to treatment not dis | sease. | | |
| CD4 count | WNL | <lln -="" 500="" mm<sup="">3</lln> | 200 - <500/mm³ | 50 - <200/mm³ | <50/mm³ |
| Haptoglobin | normal | decreased | - | absent | • |
| Hemoglobic (Hgb) | WNL | <lln -="" 10.0="" dl<br="" g=""><lln -="" 100="" g="" l<br=""><lln -="" 6.2="" l<="" mmol="" td=""><td>8.0 - &lt;10.0 g/dL<br/>80 - &lt;100 g/L<br/>4.9 - &lt;6.2 mmol/L</td><td>6.5 - &lt;\$.0 g/dL<br/>65 - &lt;80 g/L<br/>4.0 - &lt;4.9 mmol/L</td><td>&lt;6.5 g/dL<br/>&lt;65 g/L<br/>&lt;4.0 mmol/L</td></lln></lln></lln> | 8.0 - <10.0 g/dL<br>80 - <100 g/L<br>4.9 - <6.2 mmol/L | 6.5 - <\$.0 g/dL<br>65 - <80 g/L<br>4.0 - <4.9 mmol/L | <6.5 g/dL<br><65 g/L<br><4.0 mmol/L |
| For leukersis studies or bose surrow infiltratives." myelopublish processes if specified in the protocol | | 10 - C1% decrease from pretrestment | 25 -<50% decrease<br>from pretreatment | 50 -<75% doctrase<br>from protestment | |
| Hemolysis (e.g., immune<br>hemolytic anemia, drug-<br>related hemolysis, other) | BODE | only laboratory evidence of hemolysis [e.g., direct antiglobulin test (DAT, Coombs') schistocytes] | evidence of red cell<br>destruction and ≥2gm<br>decrease in hemoglobin,<br>no transfusion | requiring transfusion and/or medical intervention (e.g., steroids) | catastrophic consequences of hemolysis (e.g., recal failure, hypotension, bronchospasm, emergency spienectomy) |
| Also consider Haptoglobin, He | emoglobis. | | | | |

| | | | rade | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | , 1 | 3 | 4 |
| Leukocytes (total WBC) | WNL | <pre><lln -="" 10°="" 3.0="" 3000="" <lln="" l="" mm³<="" pre="" x=""></lln></pre> | ≥2.0 - <3.0 x 10° /L<br>≥2000 - <3000/mm³ | ≥1.0 - <2.0 x 10° /L<br>≥1000 - <2000/mm³ | <1.0 x 10° A.<br><1000/mm³ |
| For BMT studies, if specified in the protocol | WXL. | 22000 -<300 X 10°A. | 210 - 20 x 10 d<br>21000 - 20000 | - 200 x 0.7 c 2008<br>- 2000/mm² | <0.5 i 10° /L |
| Fur pediatric BMT studies<br>(using age, race and sex<br>normal values), if specified<br>in the protocol | | 25 - ZION LIN - 18 | 20 (7) UN 1 | 25-50% ILV | S28 DX |
| Lymphopenia | WNL | <lln -="" 1.0="" 10°="" l<br="" x=""><lln -="" 1000="" mm'<="" td=""><td>≥0.5 - &lt;1.0 x 10* /L<br/>≥500 - &lt;1000/mm³</td><td>&lt;0.5 x 10° /L<br/>&lt;500/mm³</td><td>•</td></lln></lln> | ≥0.5 - <1.0 x 10* /L<br>≥500 - <1000/mm³ | <0.5 x 10° /L<br><500/mm³ | • |
| For pediatric BMT studies<br>(using age, race and sex<br>normal values), if specified<br>in the protocol. | | 275 - 2100%LIN (( ) | 20) 27 SUW | SELECTION SELECT | <25%LIN |
| Neutrophils/granulocytes<br>(ANC/AGC) | WNL | ≥1.5 - <2.0 x 10° /L<br>≥1500 - <2000/mm³ | ≥1.0 - <1.5 x 10° /L<br>≥1000 - <1500/mm <sup>3</sup> | 20.5 - <1.0 x 10 /L<br>2500 - <1000/mm³ | <0.5 x 10° /L<br><500/mm <sup>3</sup> |
| For BMT studies, If specified in the protocol. | WIL TANK | ≥1 0 - <15 110° /L - <br>≥1 000 - <1500/mag* - | 203 - <1.0 × 10° /L = 205<br>≥500 - <1.000vare* | ≥0.1 - <0.5 1.10 /L<br>≥100 - <500/mm | <0.1 x 10°/L<br><1000mm* |
| For leukernik studies or home marrow infilipadive myelophihisic process, if specified in the protocol | | 10 - 23% decrease<br>from baseline | 25 - Oh screae<br>from baseline | 50 55 decrase<br from baseline | 273% decrease from<br>beacher : 1887 1987 1 |
| Platelets | WNL | <lln -="" 10°="" 75.0="" l<br="" x=""><lln -="" 75.000="" mm³<="" td=""><td>≥50.0 - &lt;75.0 x 10° /L<br/>≥50,000 - &lt;75,000/mra<sup>3</sup></td><td>≥10.0 - &lt;50.0 x 10° /L<br/>≥10,000 - &lt;50,000/mm³</td><td>&lt;10.0 x 10° /L,<br/>&lt;10,000/mm³</td></lln></lln> | ≥50.0 - <75.0 x 10° /L<br>≥50,000 - <75,000/mra <sup>3</sup> | ≥10.0 - <50.0 x 10° /L<br>≥10,000 - <50,000/mm³ | <10.0 x 10° /L,<br><10,000/mm³ |
| For BMT studies, if specified in the protocol. | WNL # | 250,000 - <75,000/mm² | ≥20,00 - <50,000 × 10° /L<br>≥20,000 - <50,000 √mm² | 210.000 20.000 TO A | 21000/em |
| For leukem's studies or bose<br>marrow infiltrative/<br>myelophthisic process. If<br>specified in the protocol. | WNL | 10 - <25% dermase<br>from beacline | 25 < 50% docresse from baseline | 50 <75% decrease<br>from baseline | 275% locrysie trons<br>basellos |
| Transfusion: Platelets | пове | | <del>-</del> | yes | platelet transfusions and<br>other measures required |
| | | | | | to improve platelet increment; platelet transfusion refractoriness associated with life-threstening bleeding. (e.g., HLA or cross matched platelet transfusions) |
| For BMT studies; if specified in the protocol. | pose | 1 piatelet transfussion in<br>24 bours | 2 placelet transfusions in<br>24 hours | 23 platelet transfusions<br>in 24 bours | platelet transfisions and other measures frautres to improve platelet increment platelet transfision |
| | rente pe gripret er be tit bie u. un | | | | with the threathing bleeding (e.g. W.A. or cross parched placed transmissions) |
| Also consider Platelets. | atter effinfflimm. De tyle et i 1920. | II var. A francis | gilli i 1944 - Sagar Aggi Melebera i Afdalama | - २ व्याप्त वर्षा स्थापति । । । १ वर्षाः ।<br>- | tallitelitelitelitelitelitelitelitelitelit |

| | | C | irade | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | . 2 | 3 | 4 |
| Transfusion: pRBCs | none | •/ | - | yes | |
| | | elective or planned | Sective or parmed | ≥4 upRBC in 24 hours | being yars associated with life threatening anemia medical |
| per flet in the products. | | SS and the process of | a norrelective or leave | | Especial required ( Especial for the second |
| | | | | | * improve hemoglobin |
| Also consider Hemoglobia. | | * | | | |
| Blood/Bone Marrow - Other (Specify,) | 000e | mild | moderate | severe | life-threatening or "disabling |
| | | CARDIOVASCUL | AR (ARRHYTHM | ſIA) | |
| Conduction abnormality/<br>Atrioventricular heart block | BORE | asymptomatic, not requiring treatment (e.g., Mobitz type I second-degree AV block, Wenckebach) | symptomatic, but not<br>requiring treatment | symptomatic and requiring treatment (e.g., Mobitz type II second-degree AV block, third-degree AV block) | life-threatening (c. g.,<br>arrhythmia associated<br>with CHF, hypotension<br>syncope, shock) |
| Nodal/junctional<br>arrbythmia/dysrbythmia | DODE | asymptomatic, not<br>requiring treatment | symptomatic, but not<br>requiring treatment | symptomatic and<br>requiring treatment | life-threatening (e.g.,<br>arrhythmia associated<br>with CHF, hypotension<br>syncope, shock) |
| Palpitations | none | present | * | • | - |
| Note: Grade palpitations only | n the absence of | a documented arrbythmia. | | | |
| Prolonged QTc interval<br>(QTc >0.48 seconds) | none | asymptomatic, not<br>requiring treatment | symptomatic, but not<br>requiring treatment | symptomatic and<br>requiring treatment | tife-threatening (e.g.,<br>ambythmia associated<br>with CHF, hypotension<br>syncope, shock) |
| Sinus bradycardia | none | asymptomatic, not<br>requiring treatment | symptomatic, but not<br>requiring treatment | symptomatic and<br>requiring treatment | life-threatening (e.g.,<br>arrhythmia associated<br>with CHF, hypotension<br>syncope, shock) |
| Sinus tachycardia | none | asymptomatic, not<br>requiring treatment | symptomatic, but not<br>requiring treatment | symptomatic and<br>requiring treatment of<br>underlying cause | - |
| Supraventricular ambythmuss<br>(SVT/atrial fibrillation/<br>flutter) | none | asymptomatic, not<br>requiring treatment | symptomatic, but not<br>requiring treatment | symptomatic and<br>requiring treatment | life-threatening (e.g.<br>arrhythrmia associated<br>with CHF, hypotension<br>syncope, shock) |
| Syncope (fainting) is graded in | the NEUROLO | GY category. | | | |
| Vasovagal episode | 2006 | - | present without loss of consciousness | present with loss of consciousness | - |

| | | Gr | nde | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | * 2 | 3 | 4 |
| Ventricular arraythmia<br>(PVCs/bigeminy/trigeminy/<br>ventricular tachycardia) | pone | equiring treatment | symptomatic, but not<br>requiring treatment | symptomatic and requiring treatment | life-threatening (e.g.,<br>arrhythmia associated<br>with CHF, hypotensio<br>syncope, shock) |
| Cardiovascular/<br>Arrhythmia - Other<br>(Specify,) | BORE | asymptomatic, not<br>requiring treatment | symptomatic, but not<br>requiring treatment | symptomatic, and<br>requiring treatment of<br>underlying cause | life-threatening (e.g.,<br>arrhythmia associated<br>with CHF, hypotensio<br>syncope, shock) |
| | | CARDIOVASCU | LAR (GENERAL | ) | |
| Acute vascular leak<br>syndrome | absent | - | symptomatic, but not<br>requiring fluid support | respiratory compromuse<br>or requiring fluids | life-threatening;<br>requiring pressor<br>support and/or<br>ventilatory support |
| Cardiac-ischemia/infarction | bone | non-specific T - wave<br>flattening or changes | asymptomatic. ST - and<br>T - wave changes<br>suggesting isothemia | angua without evidence<br>of infarction | acute myocardial<br>infarction |
| C. rdiac left ventricular<br>function | aormai | asymptomatic decline of resting ejection fraction of ≥10% but <20% of baseline value; shortening fraction ≥24% but <30% | asymptomatic but resting ejection fraction below LLN for laboratory or decline of resting ejection fraction ≥20% of baseline value; <14% shortening fraction | CHF responsive to treatment | severe or retractory<br>CHF or requiring<br>incubation |
| CNS cerebrovascular ischemi | a is graded in the | NEUROLOGY category. | | | |
| Cardiac troponis I (cTal) | normal | - | • | levels consistent with<br>unstable anging as<br>defined by the<br>manufacturer | levels consistent with<br>myocardial infarction<br>defined by the<br>manufacturer |
| Cardiac troponin T (cTnT) | aormal | ≥0.03 - <0.05 ag/mL | ≥0.05 -<0.1 ag/mL | ≥0.1 - <0.2 ng/mL | ≥0.2 ag/mL |
| Edema | aone | asymptomatic, not<br>requiring therapy | symptomatic, requiring<br>therapy | symptomatic edema<br>limiting function and<br>unresponsive to therapy<br>or requiring drug<br>discontinuation | anasarca (severe<br>generalized edema) |
| Нуреперѕіов | none | asymptomatic, transient increase by >20 mmHg (diastolic) or to >150/100° if previously WNL; not requiring treatment | recurrent or persistent or symptomatic increase by >20 mmHg (diastolic) or to >150/100* if previously WNL; not requiring treatment | requiring therapy or more intensive therapy than previously | hypertensive crisis |

| | | | Grader / | | |
|---|---|---|---|---|---|
| Adversé Event | 0 | 1 | | 3 | 4 |
| Hypotension | DOG: | changes, but not<br>requiring therepy<br>(including transse<br>orthostatic by poss | replacement or other therapy but not | requiring merapy and sustained medical artennon, but resolves without persisting physiologic consequences | sbock (a ssociated with acidemia and impeding vital organ function of to dissue hypoperfusion |
| Also consider Syncope (faint | _ | | | | |
| Notes. Allgina of Sal 15 grade | ed as Carniac-isch | emia/infarction in the CAR | DIOVASCULAR (GENERAL) | category. | |
| or three measurement | . systolic BP 65 n<br>is in 24 hours. | umHg or less in infants up t | o I year old and 70 mmHg or le | ss in children older than 1 yea | r of age, use two successin |
| Myocardids<br>- | BODE | - | * | CHF responsive to treatment | severe or refractory |
| Operative injury of vein/artery | DODE | primary sumre rep<br>for injury, but not<br>requiring transfusi | for injury, requiring | vascular occlusion<br>requiring surgery or<br>bypass for injury | myocardial infarction:<br>resection of organ (e.g<br>bowel, limb) |
| Pericardial effusion/<br>pericarditis | goge | asymptomatic effu<br>not requiring treats | | with physiologic<br>consequences | tamponade (draina ge o<br>pericardial window<br>required) |
| Peripberal arterial ischemia | none | • | brief episode of<br>ischemia managed non<br>surgically and without<br>permanent deficit | requiring surgical | life-threatening or with permanent functional deficit (e.g., amputation) |
| Phlebitis (superficial) | pone | * | present | • | _ |
| Notes: Injection site reaction i | s graded in the Di | ERNIATOLOGY/SKIN COL | egory. | | |
| | | ARDIOVASCULAR (GEN | | | |
| yncope (fainting) is graded it | | | | | |
| Thrombosis/embolism | аове | • | deep vein thrombosis,<br>not requiring<br>anticoagulant | deep vein thrombosis,<br>requiring anticoagulant<br>therapy | embolic event including pulmonary embolism |
| ein/artery operative injury is | graded as Operati | ve injury of vein/artery in t | he CARDIOVASCULAR (GEN | | |
| isceral arterial ischemia<br>1001-myocardial) | DODE | - | brief episode of isobernia managed non-<br>surgically and without permanent deficit | requiring surgical | life-threatening or with<br>permanent functional<br>deficit (e.g., resection of<br>ileum) |
| ardiovascular/<br>eneral - Other | none | mild | moderate | severe | Life-threatening or disabling |

| | | Ğr | sa: | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | .3 | 3 | 4 |
| | • * | COAGU | LATION | | |
| Note: See the HEMORRHAG | E category for grading | the seventy of blending even | its. | | |
| DIC<br>(disseminated intravascular<br>coagulation) | absent | • | • | laboratory findings<br>present with <u>no</u><br>bleeding | laboratory findings <u>and</u><br>bleading |
| Also consider Platelets. | | • | | | |
| Note: Must have increased fibe | in split products or D- | dimer in order to grade as DI | C | | |
| Fibrigogea | WNL | ≥0.75 -<1.0 x LLN | ≥0.5 - <0.75 x LLN | ≥0.25 - <0.5 x LLN | <0.25 r LLN |
| For leukenia studies or boss<br>sarrow infiltrative/<br>myelophthusic process (//<br>specified in the protocol | PYM . | 20% decrease from | 230 <40% decrease. Some protestorest value. or LLN | 240 270% decrease<br>from protestrant value<br>or LLY | |
| Partial thromboplastin time (PTT) | WNL | >ULN - SI 3 x ULN | >15-£ x ULN | >2 x ULN | - |
| Phlebitis is graded in the CAR | DIOVASCULAR (GE | NERAL) calegory. | | | |
| Prothrombia time (PT) | WNL | >ULN - \$1.5 x ULN | >1.5 - ⊈ x ULN | >2 x ULN | • |
| Thrombosis/embolism is grade | d in the CARDIOVAS | CULAR (GENERAL) careg | ory. | | |
| Thrombotic microangiopathy (e.g., thrombotic thrombocytopenic purpura/TTP or hemolytic uremic syndrome/HUS) | absent . | | | laboratory findings<br>present without clinical<br>consequences | Inboratory findings and<br>clinical consequences.<br>(e.g., CNS hemorrhage/<br>bleeding or thrombosis/<br>embolism or real<br>failure) requiring<br>therapeutic intervention |
| For BMT studies, if the state of the specified in the protocol in the protocol in the protocol in the state of the state o | | evidence of RBC destruction (schizocytosis) without relinical consequences | | evideace of RBC destruction with creatiane (>3 * ULN) act requiring dialysis | evidence of RBC in destruction; with tensi failure requires the city of the contract of the co |
| Also consider Hemoglobia, Pla<br>Note: Must have microangiopa | | smear (e.g., schistocytes, e | met cells, red cell fragments | s). | |
| Coagulation - Other<br>(Specify,) | Done | mild | moderate | severe | Life-threaterning or<br>disabling |
| | | CONSTITUTION | IAL SYMPTOMS | | |
| Fatigue<br>(lethargy, malaise, asthenia) | Dode | increased fatigue over<br>baseline, but not<br>altering normal<br>activities | moderate (e.g., decrease in performance status by 1 ECOG level or 20% Karnofsky or Lansky) or causing difficulty performing some acquires | severe (e.g., decrease in performance status by 22 ECOG levels or 40% Karoofsky or Lanky) or loss of ability to perform some activities | bedridden or dissoling |
| Note: See Appendix III for per | formance status scales. | | | | |

| | | C | rade | | -: - <del></del> |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | . 2 | 3 | 4 |
| Fever (in the absence of neutropenia, where neutropenia is defined as AGC <1.0 x 10 //L) | BOBE | 38.0 - 39.0°C (100.4 -<br>102.2°F) | 39.) -40.0°C (102.3 -<br>104.0°F) | >40.0°C (>104.0°F ) for<br><24brs | >40.0°C (>104.0°F) id<br>>24brs |
| Also consider Allergic reacti | on/hypersensitivity. | | | | |
| Note: The temperature mean. | rements listed above a | re oral or tympanic. | | | |
| Hot flashes/flushes are grade | d in the ENDOCRINE | calegory. | | | |
| Rigors, chills | Bone | mild, requiring symptomatic treatment (e.g., blanket) or son- narcotic medication | severe and/or<br>prolonged, requiring<br>narcotic medication | not responsive to<br>narcotic medication | - |
| S weating<br>(diaphoresis) | normal | mild and occasional | frequent or drenching | | - |
| Weight gain | <b>⊴</b> % | 5 - <10% | 10 - <20% | ≥20% | - |
| Also consider Ascites, Edema | L Pleural effusion (non | -malignant). | | | |
| Weight pain associated with<br>Year-Occhisive Disease (<br>(VOD) for BMT studies; if<br>specified in the protocol: | <b>25</b> | | 선 ~(03)<br>- 제1975년 - 1 | 210% or a 3 accides | 210 v.c. (Inid etention<br>Tembra in primonary<br>Enter - Sparen |
| Also consider Asciles, Edeme | Pleasi efficaco (non | -ucritaret) | | | |
| Weight loss | <5% | 5 - <10% | 10 - <20% | ≥20% | - |
| Also consider Vomiting, Deb | ydration Diarrhea. | · | | | |
| Constitutional Symptoms - Other (Specify,) | poge . | mild | moderate | severe | life-threatening or<br>disabling |
| | | DERMATO | LOGY/SKIN | | |
| Alopecia | normai | mild hair loss | pronounced hair loss | • | • |
| Bruising<br>(in absence of grade 3 or 4<br>thrombocytopenia) | Bose | localized or in<br>dependent area | generalized | • | - |
| Note: Bruising resulting from<br>HEMORRHAGE categ | grade ) or 4 thromboc<br>ory, not in the DERM | <u>vtopenia</u> is graded as Petech<br>ATOLOGY/SKIN category. | iae/purpura <u>and</u> Hemorrhag | e/bleeding with grade 3 or 4 | thrombocytopenia in the |
| Dry skia | normal | controlled with emollients | not controlled with emollients | • | ~ |
| Erythema multiforme (e.g.,<br>Stevens-Johnson syndrome,<br>toxic epidermal necrolysis) | absent | | scattered, but not<br>generalized eruption | severe or requiring IV fluids (e.g., generalized rash or painful stomattis) | life-threatening (e.g.,<br>exfoliative or electrating<br>dermatids of requiring<br>enteral or parenteral<br>nutrinonal support) |
| Flushing | absent | present | • | - | - |
| land-foot skin reaction | gone | skin changes or<br>dermatids without pain<br>(e.g., erythema, peeling) | skin changes with pain,<br>not interfering with<br>function | skin changes with pain,<br>interfering with<br>function | • |
| njection sjie reaction | Bone | pain or itching or<br>erythema | pain or swelling, with<br>inflammation or<br>phlebitis | ulceration or necrosis<br>that is severe or<br>prolonged, or requiring<br>surgery | • |
| | | Grade | | |
|---|---|---|---|---|
| 0 | 1 | •2 | 3 | 4 |
| pormal | | | - | - |
| MORRHAGE catego | ry. | | | |
| Doge | painless erythema | painful crythema | erythema with | - |
| Done | localized pigmentation changes | generalized pigmentation changes | • | _ |
| Dage | mild or localized,<br>relieved spontaneously<br>or by local measures | intense or widespread,<br>relieved spontaneously<br>or by systemic measures | intense or widespread<br>and poorly controlled<br>despite treatment | |
| ORRHAGE citegory. | | *** | | |
| Book | Laint crythems or dry desquamation | moderate to brisk erythems or a patchy moist desquaration, mostly confined to skin folds and creases; moderate adesse; moderate adesse; | confluent monst. desquimation 21.5 cm district; and not confined to skin foldes: patting oderna | skin across of ulcersion of ful inches derint may inches bleeding pot inches by miso traine or straine |
| DONE THE PROPERTY OF THE PROPE | faint crythems or dry<br>desquaration | moderate to brisk trythems or a patchy? mosts desquarantion from the mostly confined to skin folds and creases: moderate edems. | confluent moist desquarention ≥1.5 cm districter and nor continued to skin folds; pitting elemn. | st in second of full : Westellor of full : thickness derme may lacise blocking not induced by make in the property in the control of the co |
| poge | macular or papular<br>eruption or erythema<br>without associated<br>symptoms | macular or pupular eruption or erythema with pruritus or other associated symptoms covering <50% of body surface or localized desquamation or other lesions covering <50% of body surface area | symptomatic generalized erythroderma or macular, papular or vesicular eruption or desquamation covering 250% of body surface area | generalized exidiative<br>dermatitis or ulcerative<br>dermatitis |
| no is graded separatel | y as Erythema multiforme in<br>faint crythema or dry<br>desquarmation | moderate to brisk erythems or a patchy most desquamation, mostly confined to skin folds and creases; moderate edems | N category. confluent mod st designamation ≥1.5 cm diameter and no confined to skin folds: pitting oferna | skin seconds of picers-<br>tops of full thickess<br>dermic may dende<br>spouzasons beening<br>not induced by pinor |
| Noae | rescular or papular<br>eruption or erythema | macular or papular<br>cruption or crythems | symptomatic | generalized es joint ye<br>dermatits of alcests ve |
| | BORRHAGE Catego Done Done DONE DO | pormal discoloration or ridging (kolonychia) or pitting MORRHAGE category. Bone painless erythema Bone localized pigmentation changes Bone mild or localized, relieved spontaneously or by local measures DRRHAGE category. Saint crythema or dry desoparation desoparation Faint crythema or dry desoparation macular or papular eruption or erythema without associated symptoms bypersensitivity. De is graded separately as Erythema multiforme in the papular erythema or dry desoparation | anormal discoloration or indigrage (korlonychia) or putting of nail(s) or pain in nailbeds MORRHAGE category. Done painless erythema painful erythema Done localized pigmentation changes ponce mild or localized retieved spontaneously or by local measures or dry moderate to brisk desquaration crythema or a patchy mostly confined to skin oldes and creates a moderate edeans moderate edeans are patchy folds and creates a moderate or papular crythema or a dry crythema or a patchy folds and creates a patchy folds and creates a moderate edeans are proposed to a skin oldes are crythema or a dry crythema or a patchy folds and creates a patchy confined to skin folds and creates a patchy confined to skin folds and creates a patchy folds and creates a patchy confined to skin folds and creates a patchy confined to skin folds and creates a patchy confined to skin folds and creates. | pormal discoloration or ndging (Koolonychia) or patting of nail(s) or pain in nailbods MORRHAGE category. Done painless crythema painful crythema crythema with desquamation changes intense or widespread relieved spontaneously or by local measures or by systemic measures or by systemic measures. DRRHAGE crtegory. |

| | | Gr | ade , | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | <b>*2</b> | 3 | 4 |
| Urticaria<br>(hives, welts, wheals) | BORE | requinsg on medication | requiring PO or topical treatment or IV medication or steroids for <24 hours | requiring IV medication or steroids for \$24 bours | • |
| Wound-infectious | nade | cellulius | superficial infection | infection requiring IV andbiodes | necrotizing fascilitis |
| Wound-non-infectious | none | incisional separation | incisional bernia | fascial disrupood<br>withou: evisceration | fascial disruption with eviscontion |
| Dermatology/Skin - Other (Specify,) | bone | mild | moderate | severe | li fe-durent ening or<br>di sabling |
| | | _ ENDO | CRINE | | |
| Cushingoid appearance (e.g., moon face, buffalo hump, centripetal obesity, cutaneous striae) | absent | • | present | • | - |
| Also consider Hyperglycemia | | | | | |
| Feminization of male | absent | * | | present | * |
| Gyuecomastia | pone | mild | prosounced or painful | pronounced or painful<br>and requiring surgery | • |
| Hot flashes/flushes | done | mild or no more than 1<br>per day | moderate and greater<br>than I per day | - | - |
| Hypothyroidism | absent | asymptomatic,TSH<br>elevated, no therapy<br>given | symptomatic or thyroid<br>replacement treatment<br>given | patient hospitalized for manifestations of hypothyroidism | myxedema cona |
| Masculinization of female | absent | + | • | present | - |
| SIADH (syndrome of inappropriate antidiuretic bormone) | absent | • | | present | - |
| Endocrine - Other (Specify,) | noge | mild | moderate | severe | li fe-threatening or<br>disabling |
| | | GASTROIN | TESTINAL | | |
| Amylase is graded in the MET | TABOLIC/LABORAT | ORY category. | | | |
| Авогехіа | sone . | loss of appetite | oral intake significantly<br>decreased | requiring IV fluids | requiring feeding tube<br>or parenteral nutrition |
| Ascites (non-malignant) | goge . | asymptomatic | symptomatic, requiring diurencs | symptomatic, requiring<br>therapeutic paracentesis | life-threatening<br>physiologic<br>consequences |
| Colitis | none | - | abdominal pain with<br>mucus and/or blood in<br>stool | abdominal pain, fever, change in bowel habits with ileus or peritoneal signs, and radiographic or biopsy documentation | perforation or requiring surgery or toxic megacolon |
| Also consider Hemorrhage/ble<br>Rectal bleeding/hematocnezia | | 4 thrombocytopenia, Hemorr | hage/bleeding without grad | e 3 or 4 thrombocytopenia, l | Melena/GI bleeding. |
| Constipation | none | maning stool softener or dimary modification | requiring laxatives | obstitution requiring manual evacuation or enema | obstruction or toxic<br>megacolon |

| Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| Debydrauos | bone . | dry mucous membranes<br>and/or diminished skin<br>rurgor | requiring IV fluid<br>replacement (brief) | requiring IV fluid<br>replacement (sustained) | pemerynamic collapse<br>consequences requirate<br>intensive care; |
| Also consider Diarrhea, Vomi | ting. Stomatitis/pharyng | ritis (oral/pharyogeal mucos | sitis), Hypotension. | | ***** |
| Diambea<br>patients without colostomy: | BORC | increase of <4<br>stools/day over pre-<br>treatment | increase of 4-6<br>stoods/day, or nocturnal<br>stoods | increase of ≥7 stoots/day or incontinence; or need for parenteral support for dehydration | physiologic<br>consequences requiring<br>intensive care; or<br>bemodynamic collapse |
| patients with a colostomy: | BODE . | mild increase in loose,<br>watery colostomy<br>output compared with<br>pretreatment | moderate increase in<br>loose, watery colostomy<br>output compared with<br>pretreatment, but not<br>interfering with normal<br>activity | severe increase in loose, watery colostomy output compared with pretreatment, interfering with normal activity | physiologic<br>consequences, requiring<br>intensive care; or<br>bemodynamic collapse |
| a marter and a series of the contract of the c | | >500 - ≤1000mL of diarrhea/day >5 - ≤10 mL/kg of diarrhea/day thrombocytopenia, Hemorr | diarrhea/day | >1500mi. of discribed day | seers abdonned pan<br>with or without deals<br>with or without deals<br>with or without deals<br>with or without deals<br>are deals and deals are deals and deals are deals |
| Duodenal ulcer (requires radiographic or endoscopic documentation) | none | | requiring medical management or non- surgical treatment | uncontrolled by outpatient medical management; requiring hospitalization | perforation or bleeding,<br>requiring emergency<br>surgery |
| Dyspepsia/heartburn | DODE | mild | moderate | severe | |
| - / -h-h | | | | | - |
| Dysphagia, esophagitis, odynophagia (painful swallowing) | none | mild dysphagia, but can<br>eat regular diet | dysphagia, requiring<br>predominantly pureed,<br>soft, or liquid diet | dysphagia, requiring IV<br>bydration | complete obstruction<br>(cannot swallow saliva)<br>requiring enteral or<br>parenteral nutritional<br>support, or perforation |
| Dysphagia, esophagitis,<br>odygophagia (paiaful<br>swallowing) | | mild dysphagia, but can<br>eat regular diet | dysphagia, requiring predominantly pureed, soft, or liquid diet | bydration | (cannot swallow saliva)<br>requiring enteral or<br>parenteral nutritional<br>support, or perforation |
| Dysphagia, esophagitis, odynophagia (painful swallowing) Note: If the adverse event is ra Dysphagia-esophageal related to radiation | diation-relato grade <u>ei</u> | mild dysphagia, but can<br>eat regular diet<br>ther under Dysphagia-esopi<br>mild dysphagia, but can<br>ent regular diet | dysphagia, requiring predominantly pureed, soft, or liquid diet mageal related to radiation or dysphagia, requiring predominantly pureed, soft, or liquid diet | Dysphagia-pharyngeni relat Dysphagia requiring feeding tabe, IV hydration or hyperalimentation | (cannot swallow saliva) requiring enteral or parenteral nutritional support, or perforation ted to radiation. complete obstaction (cannot swallow all vi- |
| Dysphagia, esophagitis, odynophagia (painful swallowing) Note: If the adverse event is ra Dysphagia-esophageal related to radiation | diation-relate grade <u>ei</u> Bone Januaria diagnositis due to r | mild dysphagia, but can eat regular diet ther under Dysphagia-esopi mild dysphagia, but can ent regular diet | dysphagia, requiring predominantly pureed, soft, or liquid diet mageal related to radiation or dysphagia, requiring predominantly pureed, soft, or liquid diet | Dysphagia-pharyngeni relat Dysphagia requiring feeding tabe, IV hydration or hyperalimentation | (cannot swallow saliva requiring enteral or parenteral nutritional support, or perforation ted to radiation. complete observation (cannot swallow saliva swallow saliva s |
| Dysphagia, esophagitis, odynophagia (painful swallowing) Note: If the adverse event is ra Dysphagia esophageal related to radiation | diation-relate grade ei Bone stion, Mucosicis due to r city as Fistula-esophagen | mild dysphagia, but can eat regular diet ther under Dysphagia-esopi mild dysphagia, but can ent regular diet | dysphagia, requiring predominantly pureed, soft, or liquid diet magent related to radiation or dysphagia, requiring predominantly pureed, soft, or liquid diet | Dysphagia requiring feeding tube. IV hydration or hyperalimentation hyperalimentation dysphagia, requiring feeding tube. IV | (cannot swallow saliva) requiring enteral or parenteral nutritional support, or perforation ted to radiation. Complete Obstraction (cannot swalloy allva) includes a minor fraints of storation permution permution complete (cannot swalloy allva) includes a minor fraints of storation or permution includes a minor fraints of storation or permution includes a minor fraints of storation or includes a minor fraints of storation or includes a minor fraints of storation or includes a minor includes a m |
| Dysphagia, esophagitis, odynophagia (painful swallowing) Note: If the adverse event is ra Dysphagia-esophageal related to radiation Also consider Pain due to radiation Dysphagia-pharyageal related to radiation | diation-relate grade ei Bone Bone stion, Mucosicis due to r riy as Fistula-esophagen sone | mild dysphagia, but can eat regular diet ther under Dysphagia-esopi mild dysphagia, but can ent regular diet maid dysphagia, but can eat regular diet. | dysphagia, requiring predominantly pureed, soft, or liquid diet mageal related to radiation of dysphagia, requiring predominantly pureed, soft, or liquid diet months and predominantly pureed soft, or liquid diet. | Dysphagia requiring feeding tabe, IV hydration or hyperalimensation dysphagia, requiring feeding tabe, IV hydration or hyperalimensation dysphagia, requiring feeding tabe, IV hydration or hyperalimensation dispersion dispersion | (cannot swallow saliva requiring enteral or parenteral nutritional support, or perforation ted to radiation. Complete Objection (cannot swallow saliva incomplete objection saliva incomplete objecti |
| Dysphagia, esophagitis, odynophagia (painful swallowing) Note: If the adverse event is ra Dysphagia-esophageal related to radiation Also consider Pain due to radiation to radiation to radiation. | diation-relate grade ei Bone Bone stion, Mucosicis due to r riy as Fistula-esophagen sone | mild dysphagia, but can eat regular diet ther under Dysphagia-esopi mild dysphagia, but can ent regular diet maid dysphagia, but can eat regular diet. | dysphagia, requiring predominantly pureed, soft, or liquid diet mageal related to radiation of dysphagia, requiring predominantly pureed, soft, or liquid diet months and predominantly pureed soft, or liquid diet. | Dysphagia, requiring feeding tobe, IV hydration or hyperalimentation dysphagia, requiring feeding tobe, IV hyperalimentation hyperalimentation hyperalimentation feeding tobe, IV hyperalimentation dysphagia, requiring feeding tobe, IV hyperalimentation | (cannot swallow salival requiring enteral or parenteral nutritional support, or perforation ted to radiation. Complete obstructions (cannot swallow salival s |

| | | G | rioc | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | ī . | 2 | 3 | 4 |
| Fishila-poaryogeal | pone e | • | • | present | requiring surgery |
| Fistula-rectal/anal | 0000 | • | • | present | requiring surgery |
| Fiantience | peas | mild | moderate | - | - |
| Gastric ulcer<br>(requires radiographic or<br>endoscopic documentation) | BODE | - | requiring medical<br>management or non-<br>surgical treatment | bleeding without<br>perforation, uncon-<br>trolled by outpatient<br>medical management;<br>requiring hospitalization<br>or surgery | perforation or bleedin<br>requiring emergency<br>surgery |
| Also consider Hemorrhage/bl | eeding with grade 3 or | thrombocytopeaia. Hemon | bage/bleeding without grade | 3 or 4 thrombocytopenia. | |
| Gastritis<br> | oone | | requiring medical<br>management or non-<br>surgical treatment | uncontrolled by out- patient medical management; requiring bospitalization or surgery | Life-durentening bleeding, requiring emergency surgery |
| Also consider Hemorrhage/bli<br>Hematemesis is graded in the | | | hage/bleeding without grade | : 3 or 4 thrombocytopenia. | |
| Hematochezia is graded in the | <del></del> | <del></del> | | | |
| lleus (or neuroconstipation) | none none | gory 3 · Rectat bleeding/dem | | | |
| • • | | • | intermittent, not requiring intervention | requiring non-surgical | requiring surgery |
| Mouth dryness Mucositis | normal | mild | requiring intervention | | |
| Mouth dryness Mucositis Notes: Mucositis <u>not due to ra</u> (oral/pharyngeal mucos Radiation-related muco | normal diation is graded in the sitis), and Typhlitis; or to sitis is graded as Muco | GASTROINTESTINAL cate the RENAL/GENITOURINA | moderate regory for specific sites: ColinkRY category for Vaginitis. | intervention is, Esophagicis, Gastricis, Ste | omatitis/pharysgiti s |
| Mouth dryness Mucositis Notes: Mucositis not due to ra (oral/pharyugeal mucos Radiation-related mucos Mucositis due to radiation | normal diation is graded in the sitis), and Typhlitis; or to sitis is graded as Muco | GASTROINTESTINAL cate he RENAL/GENITOURIN/ sitis due to radiation. Crythens of the rouces. | requiring intervention moderate egory for specific sites: Coli ARY category for Vaginitis. patchy pendermembra- neus reaction (patches) generally \$1.5 cm m. diameter and non- contiguous); | intervention is, Esophagicis, Gastritis, So confluent pseudomeon- branous reaction [confluents patches] [confluents patches] [confluents patches] | omatitis/pharyagitis necests (a. deep. lalceation; ani/, michical |
| Mouth dryness Mucositis Notes: Mucositis not due to racon (oral/pharyugeal mucos Radiation-related mucos Mucositis due to radiation and the second | sormal diation is graded in the sitis), and Typhilitis; or to sitis is graded as Muco. Section 1. | GASTROINTESTINAL catche RENAL/GENITOURIN/ sitis due to radiation. crythems of the roucess. | requiring intervention moderate egory for specific sites: Coli LRY category for Vaginitis. petchy periodometrical active reaction (patches) generally \$1.5 cm in. distincter and non-model contiguous); distincter and non-model contiguous); all related to reaction of Dy | intervention is, Esophagids, Gastritis, State of the confluent precision in branch research from in the confluent precision in t | omatitis/pharyagitis necrois or deep Literation; poi individed |
| Mouth dryness Mucositis Notes: Mucositis not due to radio (oral/pharyngeal mucos) Radiation-related mucos Mucositis due to radiation June 1988 1988 1988 1988 1988 1988 1988 198 | sormal diation is graded in the sitis), and Typhilitis; or to sitis is graded as Muco. Section 1. | GASTROINTESTINAL catche RENAL/GENITOURIN/ sitis due to radiation. crythems of the roucess. | moderate regory for specific sites: Coli ARY category for Vaginitis. patchy pandomembra— nous reaction (patcher) generally \$1.5 cm m. diameter and non- couringsiss); | intervention is, Esophagids, Gastritis, State of the confluent precision in branch research from in the confluent precision in t | omatitis/pharysgitis necroit (or deep) Literation; mi, mchi blechi, not indices |
| Mouth dryness Mucositis Notes: Mucositis not due to rac (oral/pharyngeal mucos Radiation-related mucos Micositis due to radiation Micosit | normal diation is graded in the sitis), and Typhlitis; or our sitis is graded as Muconsider and the sitis is graded as Muconsider and the sitis is graded as Muconsider and the sitis is graded as a sitis in the si | GASTROINTESTINAL catche RENAL/GENITOURIN/ sitis due to radiation. crythems of the roucess. Crythems of the roucess. Crythems of the roucess. Crythems of the roucess. Crythems of the roucess. | moderate requiring intervention moderate regory for specific sites: Coli RY category for Vaginitis. patcay part domestic 1- patcay | confluent pseudomenn- branous reaction [confluent pseudomenn- branous reaction [confluent pseudomenn- branous reaction [confluent pseudomenn- pseudom | omatitis/pharyagitis necroit (or deep Literation; polyticals) bleeding polyticals bleeding polyticals |
| Mouth dryness Mucositis Notes: Mucositis not due to racord (oral/pharyageal mucos Radiation-related mucos Macositis due to radiation and the state of treatment. | normal diation is graded in the sitis), and Typhlitis; or to sitis is graded as Muco sitis is graded as Muco sitis is graded as Muco sitis is graded as Muco sitis is graded as sitis graded as sitis is graded as sitis graded as sit | GASTROINTESTINAL catche RENAL/GENITOURIN/ sitis due to radiation. crythems of the roucess. | moderate requiring intervention moderate regory for specific sites: Coli RY category for Vaginitis. patcay part domestic 1- patcay | intervention is, Esophagids, Gastrius, State of the confluent precision of the confluent precision of the confluent precision of the confluent patches of the confluent of the | omatitis/pharysgitis necests of deep lateration; may niche latera |

| Grace | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | | 2 | 3 | 4 |
| Procticis | pone . | increased stool frequency, occasional blood-streaked stool; or rectal discomfort (including hemorrhoods) not requiring medication | increased stool<br>frequency, biceding,<br>mucus discharge, or<br>recall discomfort<br>requiring medicanon;<br>anal fissure | increased sool frequency/diameta requiring parenteral support; rectal bleeding requiring transfusion; or persistent mucus discharge, necessitating pads | perforation, bleeding or<br>necrosis or other life-<br>threatening<br>complication requiring<br>surgical intervention<br>(e.g., colonomy) |
| | | 3 or 4 thrombocytopenia, Hemorr | hage/bleeding without grad | e 3 or 4 thrombocytopenia. | Paín due to radiation. |
| Notes: Fistula is graded sepa<br>Proctitis occurring me<br>Appendix IV) | | and/anal.<br>er the start of radiation therapy is | graded in the RTOG/EORT | C Late Radiation Morbidity | Scoring Scheme. (See |
| Salivary gland changes | Độne | slightly thickened saliva; may have slightly altered taste (e.g., metallic); additional fluids may be required | thick, ropy, sticky saliva; markedly altered taste; alteration in diet required | | acute sali vary gland<br>necrosi s |
| Sease of smell | normal | slightly altered | markedly altered | • | - |
| Stomatius/pharyngiüs<br>(oral/pharyngeal mucosiüs) | вове | painless ulcers,<br>erythema, or mild<br>soreness in the absence<br>of lesions | painful erythema,<br>edema, or ulcers, but<br>can ear or swallow | painful erythema,<br>edema, or ulcers<br>requiring IV bydration | severe ulcention or<br>requires parenteral or<br>enteral nutritional<br>support or prophylactic<br>intubation |
| Por BMT studies if specified in the protocol. | | painless ülcers, crysheurs, or mild screens in the absence of lesions | painful crythems colorie or ulcers but cas colorie or ulcers but cas colories or ul | painful crythems, ecens, or pieces, or pieces or pieces or preventing systems or position or prepared for castenal support | |
| Note: Radiation-related muco Taste disturbance (dysgeusia) | normal | slightly aftered | markedly altered | - | • |
| Typhlitis<br>(inflammation of the cecum) | вове | - | - | abdominal pain, dia. 'ea, lever, and radiographic or biopsy documentation | perforation, bleeding or necrosis or other life-threatening complication requiring surgical intervention (e.g., colosomy) |
| Also consider Hemorrhage/bl<br>neutropenia. | eeding with grade : | or 4 thrombocytopenia, Hemorrh | age/bleeding without grade | : 3 or 4 thrombocytopenia, I | Hypotension, Febrile |
| Vomiding | BORE | l episode in 24 bours<br>over pretreatment | 2-5 episodes in 24 hours<br>over pretreatment | ≥6 episodes in 24 hours<br>over pretreatment; or<br>need for IV fluids | requiring parenteral<br>nutrition; or physiologic<br>consequences requiring<br>intensive care;<br>hemodynamic collapse |
| Also consider Dehydration. | | | | | |
| Weight gain is graded in the C | | | | | |
| Weight loss is graded in the C | BODE | L SYMPTOMS category. | moderate | severe | life-threatening or |

| | | | Grade | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | . 1 | 2 | 3 | 4 |
| | | немо | ORRHAGE | | |
| Notes: Transfusion in this se | coos refers to p | RBC infusion. | | ************************************** | |
| For <u>any</u> bleeding wid<br>Transfusion: pRBCs | b grade 3 or 4 p<br>and Transfusio | latelets (<50.000), <u>siwavs</u> grade Ho<br>n: platelets in addition to grading s | emorrhage/bleeding with g<br>severity by grading the site | grade 3 or 4 thrombocytopenia. A | Uso conside Pluelers |
| If the site or type of I<br>Hematemesis, Hemor<br>bleeding/bematochez | prysis, nemorm | eding is listed, also use the grading<br>age/bleeding with surgery, Melena<br>ding. | that incorporates the site<br>Vlower GI bleeding, Peteci | of bleeding: CNS Hemorrhage/bleed | oleeding, Hemanica.<br>ing into skin), Rectal |
| lf the platelet count is<br>≥50,000, grade Hemo | s ≥50.000 and the orbage/bleeding | e site or type of bleeding is listed, without grade 3 or 4 thrombocyto | grade the specific site. If to<br>penia and specify the site | he site or type is got listed and to<br>or type in the OTHER category. | he platelet count is |
| Hemorrhage/bleeding with | <u>0</u> 000 | mild without | | requiring transfusion | catastrophic bleeding. |
| grade 3 or 4<br>thrombocytopenia | | transivuoa | | | requiring major non-<br>elective intervention |
| Also consider Platelets, Hem (Specify site,). | oglobia, Transi | usion: platelets, Transiusion: pRB | Cs. site or type of bleeding | . If the site is not listed, grade a | is Hemorria ge-Other |
| Note: This adverse event mu | । प्र be graded fo | rany bleeding with gade 3 or 4 th | rombocytopenia. | | |
| Hemorrhage/bleeding without grade 3 or 4 | none | mild without | | requiring transfusion | caustrophic bleeding |
| thrombocytopenia | | ចលរហិរណ្ឌ | | | requiring major non-<br>elective intervention |
| Also consider Platelets, Hem | oglobin. Transf | usion: platelets, Transfusion: pRBC | Cs. Hemorrhage - Other (S | pecify site | |
| Note: Bleeding in the absent<br>HEMORRHAGE cate | ce of grade 3 or<br>gory. Also grad | 4 thrombocytopenia is graded here e as Other in the HEMORRHAGE | only if the specific site of category. | type of bleeding is not listed el | sewhere in the |
| CNS bemorrhage/bleeding | BOBE | | • | bleeding noted on CT or<br>other scan with no<br>clinical consequences | bemorthagic stroke or<br>bemorthagic vascular<br>event (CVA) with<br>neurologic signs and<br>symptoms |
| Epistaxis | none | mild without<br>transfusion | | requiring transfusion | catastrophic bleeding,<br>requiring major non-<br>elective intervention |
| Hematemesis | none | mild without<br>transfusion | • | requiring transfusion | caustrophic !seding.<br>requiring major non-<br>elective intervention |
| Hematuria<br>(in the absence of vaginal<br>bleeding) | <b>300e</b> | microscopic auly | intermittent gross<br>bleeding, no clots | persistent gross bleeding or clots; may require catheterization or instrumentation, or transitision | open surgery or necrosis<br>or deep bladder<br>ulceration |
| Hemoprysis | none | mild without<br>transfusion | - | requiring transfusion | catastrophic bleeding.<br>requiring major non-<br>elective intervention |
| Hemorrhage/bleeding associated with surgery | вопе | mild without<br>transfusion | • | requiring transfusion | catastroptus bleeding.<br>requiring major non-<br>elective intervention |
| | be time of surge | ry is not graded as an adverse ever | at. | | |
| Melena/GI pleeding | soae | mild witzout<br>transfusion | • | requinas gaesiusioa | cumstornic aleeding.<br>requiring major non-<br>elective intervention |

| : | | Gr | a de | | |
|---|---|---|---|---|---|
| Adverse Event | ð | 1 | 2 | 3 | 4 |
| Petechiae purpura<br>(nemorrhage/bieeding into<br>skin or mucosa) | none ,* | rare petechase of skin | petectuae of purpura in<br>dependent areas of skin | generalized petechae or<br>purpura of skin or<br>petechiae of any<br>mucosal site | |
| Recial bleeding/<br>bematocnezia | DOBE | mild without<br>transfusion or<br>medication | persistent, requiring medication (e.g., steroid suppositories) and/or break from radiation treatment | equiriag ganstusion | cata strophic bleeding,<br>requiring major and<br>elective intervention |
| Vaginal bleeding | none | sporting, requiring <2<br>pads per day | requiring ≥2 pads per<br>day, but not requiring<br>transfusion | requiring transfusion | catastrophic bleeding.<br>requiring major non-<br>electrive intervention |
| Hemorrhage - Other (Specify site,) | nane<br>~- | mild without<br>transfusion | • | requiring transfusion | cata strophic bleeding.<br>requiring major non-<br>elective intervention |
| | | НЕРА | ATIC | | |
| Alkaline phosphatase | WNL | >ULN - 25 x ULN | >2.5 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN |
| Bilirubin | WNL | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 - 10.0 x ULN | >10.0 x ULN |
| Bilirubin associated with graft versus boat disease (GVHD) for BMT studies, if specified in the protocol. | | | ≥1 - ∞ mg/100 mL | 26 - <15 mg/100 mL | 215 ms/(00 mt |
| GGT<br>(γ - Glutamyl transpeptidase) | WNL | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN |
| Hepatic enlargement | absent | elated adverse event jochtdir | y Veno-Occlusive Disease. | Present ( ( ) ( ) ( ) ( ) | |
| Hypoalbuminemia | WNL | <ttn -="" 3="" 5="" p="" qt<=""></ttn> | 22 · <) g/dL | <2 g/dL | • |
| Liver dysfunction/ failure (clinical) | sormai | - | • | sserixis | escephalopathy or coma |
| Portal veis flow | normal | • | decreased portal vein<br>flow | reversal/retrograde<br>portal veis flow | • |
| SGOT (AST)<br>-(serum glutamic oxaloacetic<br>transaminase) | WNL | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN |
| SGPT (ALT)<br>(serum glutamic pyruvic<br>transaminase) | WNL | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN |
| Hepatic - Other (Specify,) | none | mild | moderate | severe | life-threatening or<br>disabling |
| | INF | ECTION/FEBRI | LE NEUTROPEN | VIA | |
| Catheter-related infection | gone | mild, no active<br>treatment | moderate, localized infection, requiring local or oral treatment | severe, systemic infection, requiring IV ambitions or antifuegal ceatment or mospitalization | life-threatening sepsis (e.g., septic shock) |

Grade Adverse Event 3 Febrile neutropenia DOGE Iresea Life-inreasening sepsis (fever of unknown origin (e.g., sepac speck) without clinically or microbiologically documented infection) (ANC <1.0 x 10 /L fever 238.5°C) Also consider Neutrophils Note: Hypothermia instead of fever may be associated with neutropenia and is graded here. lafection (documented Done life-threatening sepsis present clinically or (c.g., septic shock) microbiologically) with grade 3 or 4 neutropenia (ANC <1.0 x 10 /L) Also consider Neutrophils. Notes: Hypothermia instead of fever may be associated with neutropenia and is graded here. In the absence of documented infection grade 3 or 4 neutropenia with fever is graded as Febrile neutropenia. Infection with unknown bone life-directeding sepsis present ANC (e.g., septic shock) Note: This adverse event criterion is used in the rare case when ANC is unknown. Infection without попе mild, no active moderate, localized life-threatening sepsis severe, systemic acutropenia treatment infection, requiring infection, requiring [V (e.g., septic shock) local or oral treatment antibiotic or antifungal treatment, or hospitali zation Also consider Neutrophils. Wound-infectious is graded in the DERMATOLOGY/SKIN category. lafection/Febrile Bone mild moderate severe life-threatening or Neutropenia - Other disabling (Specify, LYMPHATICS Lymphatics normal mild lymphedema moderate lymphedema severe lymphedema severe lympbedema requiring compression; limiting function: limiting function with lymphocyst lymphocyst requiring ulceration antacth Lymphatics - Other none mild moderate Severe Life-threatening or (Specify, disabling METABOLIC/LABORATORY Acidosis ليستوه pH <aormal, but ≥7.3 pH <7.3 pH <7.3 with life-(metabolic or respiratory) threatening physiologic consequences Alkalosis pormal pH >normai, but ≤7.5 pH >7.5 pH >7.5 with life-(metabolic or respiratory) threatening physiologic consequences Amylase WNL >ULN - 1.5 x ULN >1.5 - 2.0 x ULN >2.0 - 5.0 x ULN >5.0 x ULN Bicarbonate WNL دلنا> - الم سقوط 11 - 15 mEa/dL 8 - 10 mEq/dL <8 mEq/dL

| | | | Grade | | - |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| CPK<br>(creatine phosphokinase) | WNL | >ULN - 2.5 x ULN | >2.5 -5 x ULN | >5 - 10 x ULN | >10 x UIN |
| Hypercalcemia | WNL | >ULN - 11.5 mg/dL<br>>ULN - 2.9 mmol/L | >11.5 - 12.5 mg/dL<br>>2.9 - 3.1 mmol/L | >12.5 - 13.5 mg/dL<br>>3.1 - 3.4 mmol/L | >13.5 mg/dL<br>Norm# 4.6< |
| Hypercholesterolemia | WNL | >ULN - 300 mg/dL<br>>ULN - 7.75 mmol/L | >300 -400 mg/dL<br>>7.75 - 10.34 mmol/L | >400 - 500 mg/dL<br>>10.34 - 12.92 mmol/L | >500 mg/dL<br>>12.92 mmol/L |
| Hyperglyœmia | WNL | >ULN - 160 mg/dL<br>>ULN - 8.9 mmol/L | >160 - 250 mg/dL<br>>8.9 - 13.9 mmol/L | >250 - 500 mg/dL<br>>13.9 - 27.8 mmol/L | >500 mg/dL<br>>27.8 mmol/L or<br>acidosis |
| Hyperkalemia | WNL | >ULN - 5.5 mmoVL | >5_5 - 6.0 mmol/L | >6.0 - 7.0 mmol/L | Nortm 0.7< |
| Hypermaguesemia | WNL | >ULN -3.0 mg/dL<br>>ULN - 1.23 mmol/L | * | >3.0 -8.0 mg/dL<br>>1.23 - 3.30 mmol/L | >8.0 mg/dL<br>>3.0 mmo/L |
| Hypernatremia | WNL | >ULN =150 mmol/L | >150 - 155 mmol/L | >155 - 160 mmol/L | >160 mmoVL |
| Hypertriglyceridemia | WNL | >ULN - 2.5 x ULN | >2.5 - \$.0 x ULN | >5.0 - 10 x ULN | >10 x ULN |
| Hyperuricemia | ₩'nL | >ULN - <10 mg/dL<br><0.59 mmoVL without<br>physiologic<br>consequences | • | >ULN - \$10 mg/dL<br>\$0.59 mmoVL with<br>physiologic<br>consequences | >10 mg/dL<br>>0.59 m.mol/L |
| Also consider Tumor lysis s | yndrome, Renai fa | lure. Creatinine, Hyperkalemia. | | | |
| Hypocalcemia | WNL | <lln -="" 8.0="" dl<br="" mg=""><lln -="" 2.0="" l<="" mmoi="" td=""><td>7.0 - &lt;8.0 mg/dL<br/>1.75 - &lt;2.0 mmol/L</td><td>6.0 - &lt;7.0 mg/dL<br/>1.5 - &lt;1.75 mmot/L</td><td>&lt;6.0 mg/dL<br/>&lt;1.5 mmol/L</td></lln></lln> | 7.0 - <8.0 mg/dL<br>1.75 - <2.0 mmol/L | 6.0 - <7.0 mg/dL<br>1.5 - <1.75 mmot/L | <6.0 mg/dL<br><1.5 mmol/L |
| Hypoglycemia | WNL | <lln -="" 55="" dl<br="" mg=""><lln -="" 3.0="" l<="" mmol="" td=""><td>40 - &lt;55 mg/dL<br/>2.2 - &lt;3.0 mmoVL</td><td>30 - &lt;40 mg/dL<br/>1.7 - &lt;2.2 mmol/L</td><td>&lt;30 mg/cIL<br/>&lt;1.7 mmol/L</td></lln></lln> | 40 - <55 mg/dL<br>2.2 - <3.0 mmoVL | 30 - <40 mg/dL<br>1.7 - <2.2 mmol/L | <30 mg/cIL<br><1.7 mmol/L |
| Hypokalemia | WNL | <lln -="" 3.0="" l<="" mmol="" td=""><td>•</td><td>2.5 - &lt;1.0 ramoVL</td><td>&lt;25 mmoVL</td></lln> | • | 2.5 - <1.0 ramoVL | <25 mmoVL |
| Hypomagnesemia | W.NL | <lln -="" 1.2="" dl<br="" mg=""><lln -="" 0.5="" l<="" mmol="" td=""><td>0.9 - &lt;1.2 mg/dL<br/>0.4 - &lt;0.5 mmoVL</td><td>0.7 - &lt;0.9 mg/dL<br/>0.3 - &lt;0.4 mmoVL</td><td>&lt;0.7 mg/dL<br/>&lt;0.3 mmo//L</td></lln></lln> | 0.9 - <1.2 mg/dL<br>0.4 - <0.5 mmoVL | 0.7 - <0.9 mg/dL<br>0.3 - <0.4 mmoVL | <0.7 mg/dL<br><0.3 mmo//L |
| Hyponatremia | WNL | <lln -="" 130="" l<="" mmol="" td=""><td>•</td><td>120 - &lt;130 mmol/L</td><td>&lt;120 mmol/L</td></lln> | • | 120 - <130 mmol/L | <120 mmol/L |
| Hypophosphatemia | WNL | <lln -3.5="" dl<br="" mg=""><lln -="" 0.8="" l<="" mmol="" td=""><td>≥2.0 - &lt;2.5 mg/dL<br/>≥0.6 - &lt;0.8 mmol/L</td><td>≥1.0 - &lt;2.0 mg/dL<br/>≥0.3 - &lt;0.6 mmol/L</td><td>&lt;1.0 mg/dL,<br/>&lt;0.1 mmol/L</td></lln></lln> | ≥2.0 - <2.5 mg/dL<br>≥0.6 - <0.8 mmol/L | ≥1.0 - <2.0 mg/dL<br>≥0.3 - <0.6 mmol/L | <1.0 mg/dL,<br><0.1 mmol/L |
| Hypothyroidism is graded in | the ENDOCRINE | category. | • | *************************************** | ····· |
| .ipase | WNL | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 - 5.0 x ULN | >5.0 x UTLN |
| Actabolic/Laboratory:-<br>Other (Specify,) | 0006 | mild | moderate | severe | Life-threatening or<br>disabling |
| | | MUSCULO | SKELETAL | | |
| arthralgia is graded in the PA | AIN category. | | | | <del></del> |
| utbritis | 800e | mild pain with inflammation, erythema or joint swelling but not interfering with function | moderate pain with inflammation, erythema, or joint sweiling interfering with function, but not interfering with activities of daily living | severe pain with inflammation. erythema, or joint swelling and interfering with activities of daily living | cti sabling |

| Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | .2 | 3 | 4 |
| Muscle weatness<br>(not due to neuropatny) | pormai | asymptomatic with weakness on physical exam | symptomane and<br>interfering with<br>function, but not<br>interfering with<br>activities of daily living | symptomatic and interfering with activities of daily living | bedridden or dissbling |
| Myalgia (tenderness or para t | a muscles) is grao | ed in the PAIN category. | | | |
| Myositis<br>(inflammation/damage of<br>muscle) | DODE | mild pain, not<br>interfering with<br>function | pain interfering with<br>function, but not<br>interfering with<br>activities of daily living | pain interfering with<br>function and interfering<br>with activities of daily<br>living | bedridden or disabling |
| Also consider CPK. | No. of | | | | _ |
| Note: Myositis implies muscl | e damage (i.e., ele | vated CPK). | | | |
| Osteodecrosis<br>(avascular necrosis) | none | asymptomatic and<br>detected by imaging<br>only | symptomatic and interfering with function, but not interfering with activities of daily living | symptomatic and<br>interfering with<br>activities of daily living | symptomatic; or<br>disabling |
| Musculoskeletal - Other (Specify,) | none | mild | moderate | severe | life-threatening or<br>disabling |
| Aphasia, recentive and/or exp | ressive is ornded: | NEURO | | | |
| Arachaoiditis/metragismus/<br>radiculitis | absent | mild pain not interfering<br>with function | moderate pain interfering with function, but not interfering with activities of daily living | severe pain interfering<br>with activities of daily<br>living | unable to function or<br>perform activities of<br>daily living; bedridder<br>paraplegia |
| Also consider Headache, Von | niting, Fever. | | | | |
| Ataxia (incoordination) | normal | asymptomatic but<br>abnormal on physical<br>exam, and not<br>interfering with<br>function | mild symptoms interfering with function, but not interfering with activities of daily living | moderate symptoms<br>interfering with<br>activities of daily living | bedridden or disabling |
| CNS cerebrovascular<br>ischemia | none | • | - | transient ischemic event<br>or attack (TLA) | permanent event (e.g.,<br>cerebral va scular<br>accident) |
| CNS hemorrhage/bleeding is | graded in the HEM | ORRHAGE category. | | | |
| Cognitive disturbances<br>carning problems | Aone | cognitive disabilive not<br>interfering with work/school | cognitive disability:<br>interfering with work/school with | cogninie disability;<br>resulting is significant<br>mipagnesi o | e en interes en |
| | | perfurmance: preservation of intelligence | performance; decline of<br>I SD (Standard<br>Deviation) or last of<br>developmental | workSchool Teaming performance; cognitive declies > 7 SD | riski<br>Nasiski i det<br>Nasiski i det |

| | ~· | | | | |
|---|---|---|---|---|---|
| | • | G. | race<br>, | | |
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| Confusion | nortnai | confusion or association or an amount and deficit of orief ouration; resolves spontaneously with no sequelae | confusion or disorientation or attention deficit interfering with fusicion, but not interfering with activities of daily living | confusion or delinum interfering with activities of daily living | harmful to others or<br>self; requiring<br>bospitalization |
| Cranial neuropathy is graded | in the NEUROLO | XXY category as Neuropathy-crani | ial. · | | |
| Delusions | normal | • | • | present | toxic psychosis |
| Depressed level of consciousness | <br>portial | somnolence or sedation<br>not interfering with<br>function | sommolence or sedation interfering with function; but not interfering with activities of daily living | obtundation or stupor;<br>difficult to arouse;<br>interfering with<br>activities of daily living | com.a |
| Note: Syncope (fainting) is g | raded in the NEUF | ROLOGY category. | | | |
| Dizziness-lightheadeduess | noge | pox interfering with<br>function | interfering with<br>function, but not<br>interfering with<br>activities of daily living | interfering with<br>activities of daily living | bedridden or disabling |
| Dysphasia, receptive and/or e | xpressive, is grade | ed under Speech impairment in the | NEUROLOGY category. | | |
| Extrapyramidal/ involuntary movement/ restlessness | noue | mild involuntary<br>movements not<br>interfering with<br>function | moderate involuntary<br>movements interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe involuntary<br>movements or torticollis<br>interfering with<br>activities of daily living | bedridden or disabling |
| Hallucinations | normal | • | • | present | toxic psychosis |
| Headache is graded in th PA | IN category. | | | | |
| <u> Lasomaia</u> | aormai | oceasional difficulty<br>sleeping not interfering<br>with function | difficulty sleeping interfering with function, but not interfering with activities of daily living | frequent difficulty<br>sleeping, interfering<br>with activities of daily<br>living | - |
| Note: This adverse event is gr | raded when insome | aia is related to treatment. If pain o | or other symptoms interfere | with sleep do NOT grade as | insomnia. |
| Irritability<br>(children <3 years of age) | normal | mild: easily consolable | moderale; requiring<br>increased attention | severe; inconsolable | of the second se |
| Leukoencephalopathy<br>associated radiological<br>findings | noae | mild increase in SAS (subarachnoid space) and/or mild ventriculomegaly; and/or small (+/- multiple) focal T2 byperintensities, involving periventricular white manter or <1/3 of susceptible areas of cerebrum | moderate increase in SAS; and/or moderate ventriculomegaly; and/or focal T2 byperintensities extending into centrum ovale; or involving 1/3 to 2/3 of susceptible areas of cerebrum | severe increase in SAS;<br>severe<br>ventriculomegaly; near<br>total white matter T2<br>byperintensities or<br>diffuse low attenuation<br>(CT); focal white matter<br>necrosis (cystic) | severe increase in SAS: severe ventriculomegaly; diffuse low attenuation with calcification (CT); diffuse white matter necrosis (MRI) |
| Memory loss | normal | memory loss not<br>interfering with<br>function | memory loss interfering<br>with function, but not<br>interfering with<br>activities of daily living | memory loss interfering<br>with activities of daily<br>living | amnesia |

| | | G | rade | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | . 2 | 3 | 4 |
| Mood alteration-anxiety, agitation | sormal . | mild mood alteration<br>not interfering with<br>function | moderate mood alteration interfering with function, but not interfering with activities of daily living | severe mood atteration interfering with accurates of daily living | ड्यांवर्की (विद्यवस्य or<br>विकादः १० ड्यी |
| Mood alteration-depression | normal | mild mood alteration<br>not interfering with<br>function | moderate mood alteration interfering with function, but not interfering with activities of daily living | severe mood alteration interfering with activities of daily living | suicidal ideaton or<br>danger to self |
| Mood alteration-eupboria | normal | mild mood alteration<br>not interfering with<br>function | moderate mood alteration interfering with function, but not interfering with activities of daily living | severe mood alteration interfering with activities of duity living | danger (o sell |
| Neuropathic pain is graded in | the PAIN category. | | - | | |
| Neuropathy-cranial | absent | - | present, not interfering<br>with activities of daily<br>living | present, interfering with activities of duly living | tife-threatening.<br>disabling |
| Neuroраthy-токог | normal | subjective weakness but<br>no objective findings | mild objective weakness interfering with function, but not interfering with activities of daily living | objective weakness<br>interfering with<br>activities of daily living | paralysis |
| Neuropathy-sensory | BOLUTA | loss of deep tendon<br>reflexes or paresthesia<br>(including tingling) but<br>not interfering with<br>function | objective sensory loss or paresthesia (including tingling), interfering with function, but not interfering with activities of daily living | sensory loss or<br>paresthesia interfering<br>with activities of daily<br>living | permanent seasory los<br>that interferes with<br>function |
| Nystagmus | absent | present | • | - | - |
| Also consider Vision-double v | isioa. | | | | |
| Personality/behavioral | normal | change, but not<br>disruptive to patient or<br>family | disruptive to patient or family | disruptive to patient and<br>family: requiring mental<br>bealth intervention | barmful to others or<br>self; requiring<br>bospitalization |
| Pyramidal tract dysfunction e.g., T tone, hyperreflexia, positive Babinski, 1 fine notor coordination) | normal | asymptomatic with abnormality on physical examination | symptomatic or interfering with function but not interfering with activities of daily living | interlering with<br>activities of daily living | bedridden or disabling<br>paralysis |
| cizue(s) | BODE | • | seizure(s) self-limited<br>and consciousness is<br>preserved | seizure(s) in which<br>consciousness is altered | seizures of any type which are prolonged, repetitive, or difficult to courd (e.g., sarus epilepticus, intractable epilepsy) |
| peech impairment<br>.g., dysphasia or aphasia) | nomal | • | awareness of receptive<br>or expressive dysphasia,<br>not impairing ability to<br>communicate | receptive or expressive<br>dysphasia, impairing<br>ability to communicate | inability to<br>communicate |
| yncope (fainting) | absent | | | present | |

| | | • | Grade 🔧 | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | . 1 | 2 | 3 | 4 |
| Tremor | BODE | mild and brief or<br>intermittent but not<br>interfering with<br>function | moderate tremor interfering with function, but not interfering with activities of daily living | severe tremor interfenog with activities of daily living | - |
| Vertigo | noue | not interfering with<br>function | interfering with<br>function, but not<br>interfering with<br>activities of daily living | interfering with activities of daily living | bedridden or disablin |
| Neurology - Other<br>(Specify,) | DODE | mild<br>—— | moderate | severe | life-threatening or<br>disabling |
| | | OCULA | R/VISUAL | | |
| Cataract | BORÉ | asymptomatic | symptomatic, partial<br>visual loss | symptomatic, visual loss requiring treatment or interfering with function | ▼ (m) |
| Conjuncti viti s | aoot | abnormal ophthalmologic changes, but asymptomatic or symptomatic without visual impairment (i.e., pain and irritation) | symptomatic and interfering with function, but not interfering with activities of daily living | symptomatic and interfering with activities of ctally living | • |
| Ory eye | normal | mild, not requiring treatment | moderate or requiring | * | • |
| Glaucoma | DODE | increase in intraocular<br>pressure but no visual<br>loss | increase in intraocular<br>pressure with retinal<br>changes | visual impairment | unilateral or bilateral<br>loss of vision<br>(blindness) |
| Ceratitis<br>comeal inflammation/<br>orneal ulceration) | no ac | abuormal ophthalmologic changes but asymptomatic or symptomatic without visual impairment (i.e., pain and irritation) | symptomatic and interfering with function, but not interfering with activities of daily living | symptomatic and interfering with activities of daily living | unilateral or bibleral<br>loss of vision<br>(blindness) |
| earing (watery eyes) | BODE | mild: not inter <u>fering</u><br>with function | moderate: interfering with function, but not interfering with activities of daily living | interfering with<br>activities of daily living | • |
| ision-blurred vision | BOTMal | - | symptomatic and interfering with function, but not interfering with activities of daily living | symptomatic and interfering with activities of daily living | - |
| sion-double vision<br>plopia) | normal | • | symptomatic and interfering with function, but not interfering with activities of daily living | symptomatic and interfering with activities of daily living | |
| sion-flashing<br>1 | normal | mild, not interfering<br>with function | symptomatic and interfering with function, but not interfering with activities of daily living | symptomatic and interfering with activities of daily living | - |

70

| Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | •2 | 3 | 4 |
| Vision-aight blindness<br>(nyctalopia) | BOLUTI | abnormal electro-<br>reunography but<br>asymptomatic | symptomadic and interferog with interferog with according with according to faily living | symptomatic and<br>interfering with<br>activities of duly living | - |
| Vision-photophobia | BOCHEJ | • | symptomatic and interiering with function, but not interfering with activities of daily living | symptomatic and interfering with activities of daily living | - |
| Ocular/Visual - Other<br>(Specify,) | oormal | mild | moderate | Severe | unilateral or bilateral<br>loss of vision<br>(blindness). |
| | | PA | LIN | | - |
| Abdomiaal pain or cramping | aoae | mild pain not interfering<br>with function | moderate pain: pain or<br>analgesics interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe pain: pain or<br>analgesics severely<br>interfering with<br>activities of daily living | di sabling |
| Arthralgia<br>(joint pain) | none | mild pain not interfering<br>with function | moderate pain: pain or<br>analgesics interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe pain: pain or<br>analgesics severely<br>interfering with<br>activities of daily living | disabling |
| Arthrids (joint pain with clinic | al signs of inflam | mation) is graded in the MUSCU | LOSKELETAL category. | | |
| Bone pain | uone | mild pain not interfering<br>with function | moderate pain: pain or<br>analgesics interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe pain: pain or<br>analgesics severely<br>interfering with<br>activities of daily living | disabling |
| Chest pain<br>(non-cardiac and non-<br>pleuritic) | gode | mild pain not interfering<br>with function | moderate pain: pain or<br>analgesics interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe pain: pain or<br>analgesics severely<br>interfering with<br>activities of daily living | disabling |
| Dysmeporrbea | none | mild pain not interfering<br>with function | moderate pain: pain or<br>analgesics interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe pain: pain or<br>analgesics severely<br>interfering with<br>activities of daily living | disabling |
| Dyspareunia | sose | mild pain not interfering<br>with function | moderate pain<br>interfering with sexual<br>activity | severe pain preventing<br>sexual activity | • |
| Dysuria is graded in the RENA | ALJGENTTOURD | NARY category. | | | |
| Earache (otalgia) | none | mild pain not interfering<br>with function | moderate pain: pain or<br>analgesics interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe pain: pain or<br>analgesics severely<br>interfering with<br>activities of daily living | disabling |
| Headache 1 | none | mild pain not interfering<br>with function | moderate pain: pain or<br>analgesics interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe pain: pain or<br>analgesics severely<br>interfering with<br>activities of daily living | disabli a g |

| Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | .2 / | 3 | ٤ |
| Hepatic pain | pose | muld pain not intervening<br>with function | moderate odus: peus or<br>analgesics interiering<br>with function, but not<br>interfering with<br>activities of daily living | severe puin: pain or<br>analgesics severely<br>interiering with<br>activities of daily living | di sebuag |
| Myaigia<br>(muscle pain) | BODE | mild pain not interfering<br>with function | moderate pain; pain or<br>analgesics interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe pain: pain or<br>enalgesics severely<br>interfering with<br>activities of daily living | dissibling |
| Neuropathic pain<br>(e.g., jaw pain, neurologic<br>pain, phantom limb pain,<br>post-infectious neuralgia, or<br>painful neuropathies) | DODE . | mild pain not interfering<br>with function | moderate pain; pain or<br>analgesics interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe pain: pain or<br>analgesics severely<br>interfering with<br>- activities of daily living | disabling |
| Pain due to radiation | Philippia Control (see 40) | mild pain not interfering<br>with fraction | moderate para: para or<br>anxigency interfering !<br>with function, but not<br>interfering with """<br>activities of daily living | sever: paint pain of analycises severely interfering with activities of daily hiving | disabling |
| Pelvic pain | Bone | mild pain not interfering<br>with function | moderate pain: pain or<br>analgesics interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe pain: pain or<br>analgesics severely<br>interfering with<br>activities of daily living | disabling |
| Pleuritic pais | sone | mild pain not interfering<br>with function | moderate pain: pain or<br>analgesics interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe pain: pain or<br>analgesics severely<br>interfering with<br>activities of daily living | disabling |
| Rectal or perirectal pain<br>(proctalgia) | рове | mild pain not interfering<br>with function | moderate pain: pain or<br>analgesics interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe pain: pain or<br>analgesics severely<br>interfering with<br>activities of daily living | disabling |
| Tumor pain<br>(onset or exacerbation of<br>tumor pain due to treatment) | none | mild pain not interfering<br>with function | moderate pain: pain or<br>analgesics interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe pain: pain or<br>anal <sub>b</sub> usics severely<br>interfering with<br>activities of daily living | disabling |
| Tumor flare is graded in the SY. | NDROME category. | | <u></u> | | |
| Pais - Other<br>(Specify,) | none . | mild | moderate | severe | disabling |
| | | PULMO | NARY | | |
| Adult Respiratory Discress | absent | • | - | - | present |
| Syndrome (ARDS) | | | | | |

| Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | .2 | 3 | 4 |
| Carbon monoxide diffusion capacity (DL <sub>CO</sub> ) | 290% of<br>pretreatment or ."<br>normal value | ≥75 - <90% of<br>protreatment or normal<br>value | ≥50 - <75% of pretreatment or normal value | ≥25 - <50% of<br>I pretreatment or normal<br>value | 25% of pretratment<br>or normal value |
| Cough | absent | mild, relieved by pon-<br>prescription medication | requiring narcotic<br>antitussive | severe cough or coughing spasms, poorly controlled or unresponsive to treatment | • |
| Dyspnea<br>(shortness of breath) | вогтыі | • | dyspaca da exemioa | dyspnea at normal level<br>of activity | entition senginor dashers at teator |
| FEV, | 290% of pretreatment or normal-value | ≥75 -<90% of pretreatment or normal value | ≥50 - <75% of pretreatment or normal value | ≥25 -<50% of<br>pretreatment or normal<br>value | 25% of pretreatment or normal value |
| Hiccoughs (hiccups, singultus) | DODE | mild, not requiring<br>treatment | moderate, requiring<br>treatment | severe, prolonged, and<br>refractory to treatment | - |
| Нурохіа | normal | - | decreased O2 saturation with exercise | decreased O <sub>3</sub> saturation<br>at rest, requiring<br>supplemental oxygen | decressed O: situration requiring pressure support (CPAP) or assisted ventilation |
| Pleural effusion<br>(non-malignant) | BODE | asymptomatic and not<br>requiring creatment | symptomatic, requiring<br>diuretics | symptomatic, requiring O2 or therapeutic thoraceutesis | li fe-threatening (e.g.,<br>requiring intubation) |
| Pleuritic pain is graded in the l | PAIN category. | | | | |
| Facumonitis/pulmonary<br>infiltrates | pone . | radiographic changes<br>but asymptomatic or<br>symptoms not requiring<br>steroids | radiographic changes<br>and requiring steroids of<br>diuretics | radiographic changes<br>or and requiring oxygen | radiographic changes<br>and requiring assisted<br>ventilation |
| Pseumothorax . | DOBE | no intervention required | chest tube required | sclerosis or surgery required | li fe-threatening |
| Pulmonary embolism is graded | as Thrombosis/embol | ism in the CARDIOVASCU | LAR (GENERAL) categ | ory. | |
| Pulmonary fibrosis | gone | radiographic changes,<br>but asymptomatic or<br>symptoms not requiring<br>steroids | requiring steroids or<br>diuretics | requiring oxygen | requiring assisted<br>ventilation |
| Note: Radiation-related pulmos | ary librosis is graded | in the RTOG/EORTC Late R | adiation Morbidity Scor | ing Scheme-Lung. (See Appea | dix IV) |
| Voice changes/stridor/larynx<br>e.g., hoarseness, loss of<br>voice, laryngitis) | normal | mild or interminent<br>boarseness | persistent boarseness,<br>but able to vocalize;<br>may have mild to<br>moderate edema | whispered speech, not<br>able to vocalize; may<br>have marked edema | marked dy spued/stri do<br>requiring trachestomy<br>or intubation |
| Notes: Cough from radiation is | graded as cough in the | PULMONARY category. | | | |
| Radiation-related bemop<br>related bemoptysis from | etysis from larynx/phar<br>the thoracic cavity is ; | rynx is graded as Grade 4 M<br>graded as Grade 4 Hemopty | ucositis due to radiation<br>sis in the HEMORRHA( | in the GASTROINTESTINAL<br>GE category. | category. Radiation- |
| ulmonary - Other<br>Specify,) | none | mild | moderate | severe | li fe-threatening or<br>di sabling |

| | Grade | | | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | • 2 | 3 | 4 |
| | e/<br> | RENAL/GEN | NITOURINARY | | |
| Bladge: spasms | abseni | mild symptoms, not<br>requiring intervention | symptoms requiring antispasmodic | severe symptoms<br>requiring narcotic | * |
| Creatinine | WNL | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 - 6.0 x ULN | >6.0 ± ULN |
| Note: Adjust to age-appropri | iate levels for pediatric | грапени. | | | |
| Dysuria<br>(psiaful urination) | none | mild symptoms<br>requiring no<br>intervention | symptoms relieved with<br>therapy | symptoms not relieved<br>despite therapy | |
| Figula or GU fistula<br>(e.g., vaginal, vesicovaginal) | bone | • | • | requiring intervention | requiring surgery |
| Hemoglobinurii | * | present | • | • | • - |
| Hemanuria (in the absence of | vaginal bleeding) is gr | aded in the HEMORRHAGE | category. | | |
| Incontinence | none | with coughing,<br>sneezing, etc. | spontaneous, some control | ao control (in the<br>absence of fistula) | • |
| Operative injury to bladder<br>and/or ureter | вове | - | injury of bladder with<br>primary repair | sepsis, fistula, or obstruction requiring secondary surgery; loss of one kidney; injury requiring anastomosis or re-implantation | septic obstruction of<br>both kidneys or<br>vesicovaginal fistula<br>requiring diversion |
| Proteinuria | normal or <0.15<br>g/24 hours | 1+ or 0.15 - 1.0 g/24<br>bours | 2+ to 3+ or 1.0 - 3.5<br>g/24 hours | 4+ or >3.5 g/24 bours | nephrotic syndrome |
| Note: If there is an inconsister | scy between absolute v | alue and dip stick reading, u | se the absolute value for grad | ding. | |
| Regal failure | none | • | • | requiring dialysis, but<br>reversible | requiring dialysis and<br>irreversible |
| Ureteral obstruction | Done | unilateral, not requiring surgery | - | bilateral, not requiring surgery | steat aephrosomy |
| Unnary electrolyte wasting<br>(e.g., Fanconi's syndrome,<br>maal tubular acidosis) | Bone | asymptomatic, not<br>requiring treatment | mild. reversible and<br>manageable with oral<br>replacement | reversible but requiring<br>IV replacement | irreversible, requiring continued replacemen |
| Also consider Acidosis, Bicarl | bonate, Hypocalcemia, | Hypophosphatem1. | | | |
| Jrinary frequency/urgency | normal | increase in frequency or<br>nocturia up to 2 x<br>normal | increase >2 x normal<br>but<br>bourly | bourly or more with urgency, or requiring catheter | ************************************** |
| Trinary retention | oormal | besitancy or dribbling,<br>but no significant<br>residual urine; retention<br>occurring during the<br>immediate<br>postoperative period | besitancy requiring medication or occasional in/out catheterization (<4 x per week), or operative bladder atony requiring indwelling catheter beyond immediate postoperative period but for <6 weeks | requiring frequent in/out catheterization (24 x per week) or urological intervention (e.g., TURP, suprapublic tube, urethrotomy) | bladder ru prure |





| | Grade | | | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| Autoimmune reactions a | Autoimmune reactions are graded in the ALLERGY/CMMUNOLOGY category. | | | | |
| DIC (disseminated intrav | DIC (disseminated intravascular congulation) is graded in the COAGULATION entegory. | | | | |
| Fan∞ni's syndrome is g | raded as Urinary elect | rolyte waxing in the RENALIGE | TTOURINARY category. | | |
| | ······································ | ectrolyte wasting in the RENAL/GI | | | |
| | | me) is graded in the DERMATOL | | | |
| | | c hormone) is graded in the ENDO | <del></del> | | |
| | | thrombocytopenic purpura/TTP or | | e/HUS) is ended in the CO | AGI II ATION |
| Tumor flare | BORE | mild pain sot intertering<br>with function | moderate pain; pain or<br>analgesics interfering<br>with function, but not<br>interfering with<br>activities of daily living | severe pain: pain or analgesics interfering with function and interfering with activities of daily living | Disabling . |
| Also consider Hypercalce | mia. | | | | |
| Note: Tumor flare is char<br>hormones). The sy | racterized by a conste<br>mptoms/signs include | llation of symptoms and signs in d<br>tumor pain, inflammation of visib | irect relation to initiation of<br>de turnor, hypercalcemia, di | therapy (e.g., anti-estrogen<br>(fuse bone pain, and other e | vandrogens or additional<br>lectrolyte disturbances. |
| Tumor tysis syndrome | absent | • | | present | • |
| Also consider Hyperkalen | nia, Creatinine. | | | | |
| Urinary electrolyte wastin | Urinary electrolyte wasting (e.g., Fanconi's syndrome, renal tubular acidosis) is graded in the RENAL/GENITOURINARY category. | | | | |
| Syndromes - Other (Specify,) | pone | mild | moderate | severe | life-threatening or<br>disabling |

### Adverse Event Modulé

To be implemented at the request of the study sponsor or principal investigator in the protocol or by protocol amendment when more detailed information is considered pertinent.

| Adverse Event: | Date of Treatment: | | Course Numb | er: | |
|---|---|---|---|---|---|
| Date of onset: | | | Grade at onse | t: | |
| Date of first change in grade: | | | Grade: | | |
| Date of next change in grade: | | | Grade: | | |
| Date of next change in grade: | | **** | Grade: | | |
| Date of next change in grade: | The Part | | Grade: | | |
| Date of next change in grade: | | | Grade: | | |
| Date of next change in grade: | | | Grade: | | |
| Did adverse event resolve? If so, date of resolution of adverse event: | Ycs | No | | | <del></del> |
| Date of last observation (if prior to recovery): | | | | | ······································ |
| Reason(s) observations stopped (if prior to recovery): | | | | | |
| Was patient retreated? | Yes | No | | <u> </u> | |
| If yes, was treatment delayed for recovery? | Yes | No | | | |
| Date of next treatment? | 1 03 | 110 | | | |
| Dose reduced for next treatment? | Yes | No | | | |
| Additional Comments: | | | | | |
| If module is being activated for new adverse Grade 0 = | | | | ad verse event grading | <b>g</b> : |
| Grade = | | | | _ | |
| Grade 2 = | | | | <u>.</u> | |
| Grade 3 = | | | | _ | |
| Grade 4 = | | | | | |

# Infection Module

To be implemented at the request of the study sponsor or principal investigator in the protocol or by protocol amendment when more detailed information is considered pertinent.

| 1. | Use the Common | Poxicity Criteria | definitions to grade | the severity of the in | fection. |
|---|---|---|---|---|---|
| 2. | Specify type of inf | ection from the f | ollowing (CHOOSE | ONE): | |
| | BACTERIAL | FUNGAL | PROTOZOAL | VIRAL | UNKNOWN |
| 3. | Specify site of infe | ction from the fo | llowing (CHOOSE | ALL THAT APPLY | ): |
| | BLOOD CULTUR<br>BONE INFECTIO<br>CATHETER (intra<br>CATHETER (intra<br>CENTRAL NERV<br>EAR INFECTION<br>EYE INFECTION<br>GASTROINTEST!<br>ORAL INFECTION<br>PNEUMONIA<br>SKIN INFECTION<br>UPPER RESPIRAT<br>URINARY TRACT | E POSITIVE N venous) venous), tunnel i OUS SYSTEM I INAL INFECTION I TORY INFECTION TION | nfection<br>NFECTION | | |
| 4. | Specify organism, i | f known: | * | | |
| 5. | Prophylactic antibio | otic, antifungal, c | or antiviral therapy a | dministration | |
| | Yes 1 | No | | | |
| | If prophylaxis was | given prior to inf | ection, please specil | y below: | |
| | Antibiotic prophyla | xis | | | |
| | Antifungal prophyla | axis | | | Market and the state of the sta |

# Performance Status Scales/Scores

# PERFORMANCE STATUS CRITERIA

| | ECOG (Zubrod) | | Karnofsky | Karnotsky Lansky* | |
|---|---|---|---|---|---|
| Score | Description | Score | Description | Score | Description |
| 0 | G Fully active, able to carry on | | Normal, no complaints, no evidence of disease. | 100 | Fully active, normal. |
| | all pre-disease performance without restriction. | 90 | Able to carry on normal activity; minor signs or symptoms of disease. | 90 | Minor restrictions in physically strenuous activity. |
| 1 | Restricted in physically atrenuous activity but | 80 | Normal activity with effort;<br>some signs or symptoms of<br>disease. | 80 | Active, but tires more quickly |
| | ambulatory and able to carry<br>out work of a light or<br>sedentary nature, e.g., light<br>housework, office work. | 70 | Cares for self, unable to carry on normal activity or do active work. | 70 | Both greater restriction of and less time spent in play activity. |
| 2 | Ambulatory and capable of all selfcare but unable to carry | 60 | Requires occasional assistance, but is able to care for most of his/her needs. | 60 | Up and around, but minimal active play, keeps busy with quieter activities. |
| | out any work activities. Up<br>and about more than 50% of<br>waking hours. | 50 | Requires considerable assistance and frequent medical care. | 50 | Gets dressed, but lies around much of<br>the day; no active play; able to<br>participate in all quiet play and<br>activities. |
| 3 | Capable of only limited selfcare, confined to bed or | 40 | Disabled, requires special care and assistance. | 40 | Mostly in bed; participates in quiet activities. |
| | chair more than 50% of waking hours. | _ 30 | Severely disabled,<br>hospitalization indicated.<br>Death not imminent. | 30 | In bed; needs assistance even for quiet play. |
| 4 | Completely disabled. Cannot carry on any selfcare. Totally | 20 | Very sick, hospitalization indicated. Death not imminent. | 20 | Often sleeping; play entirely limited to very passive activities. |
| | confined to bed or chair. | 10 | Moribund, fatal processes progressing rapidly. | 10 | No play; does not get out of bed. |

<sup>\*</sup>The conversion of the Lansky to ECOG scales is intended for NCI reporting purposes only.

# RTOG/EORTC Late Radiation Morbidity Scoring Scheme Use for adverse event occurring greater than 90 days after radiation therapy.

| Crade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| Bladder-<br>Late RT Morbidity Scoring | No change from<br>baseline | Slight epithelial<br>atrophy/minor<br>telangiectasia<br>(microscopic hematuria) | Moderate frequency/<br>generalized<br>telangiectasia/<br>intermittent<br>macroscopic hematuria | Severe frequency and dysurial severe generalized telangicetasia (often with petechiae); frequent hermaturia; reduction in bladder capacity (<150 mL) | Necrosis/contracted<br>bladder (capacity <100<br>mL)/severe<br>bemorrhagic cystitis |
| Bone-<br>Late RT Morbidity Scoring | No change from<br>baseline | Asymptomatic; no growth retardation; reduced bone density | Moderate pain or<br>tenderness; growth<br>retardation; irregular<br>bone sclerosis | Severe pain or tenderness; complete arrest of bone growth; dense bone selerosis | Necrosis/<br>spontateous fracture |
| Brain-<br>Late RT Morbidity Scoring | No change from<br>baseline | Mild beadache: slight<br>lethargy | Moderate beadache;<br>great lethargy | Severe headaches;<br>severe CNS dysfunction<br>(partial loss of power or<br>dyskinesia) | Seizures or paralysis;<br>coma |
| Esophagus-<br>Late RT Morbidity Scoring | No change from<br>baseline | Mild librosis; slight<br>difficulty in swallowing<br>solids; no pain on<br>swallowing | Unable to take solid food normally; swallowing semi-solid food; dilation may be indicated | Severe fibrosis; able to<br>swallow only liquids;<br>may bave pain on<br>swallowing; dilation<br>required | Necrosis/<br>perforation: fistula |
| Eye-<br>Late RT Morbidity Scoring | No change from<br>baseline | Asymptomatic cataract;<br>minor corneal<br>ulceration or keratitis | Symptomatic estaract:<br>moderate corneal<br>ulceration; minor<br>recinopathy or glaucoma | Severe keratitis; severe retiaopathy or detachment; severe giaucoma | Panophthalmitis;<br>blindness |
| Heart-<br>Late RT Morbidity Scoring | No change from<br>baseline | Asymptomatic or mild symptoms: transient T wave inversion and ST changes; sinus tachycardia > 1 10 (at rest) | Moderate angina on effort; mild pericarditis; normal heart size; persistent abnormal T wave and ST changes; low QRS | Severe angina; pericardial effusion; constrictive pericarditis; moderate beart failure; cardiac enlargement; EKG abnormalities | Tamponade/severe beart<br>failure/severe<br>constrictive pericarditis |
| loint-<br>Late RT Morbidity Scoring | No change from baseline | Mild joint stiffness;<br>slight limitation of<br>movement | Moderate stiffness;<br>intermittent or moderate<br>joint pain; moderate<br>limitation of movement | Severe joint stiffness;<br>pain with severe<br>limitation of movement | Necrosis/complete fixation |
| Kidney-<br>Late RT Morbidity Scoring | No change from<br>baseline | Transient albuminuma: no hypertension; mild impairment of renal function; urea 25 - 35 mg%; creatinine 1.5 - 2.0 mg%; creatinine clearance >75% | Persistent moderate albuminuria (2+); mild bypertension; no related anemia; moderate impairment of renal function; urea >36 - 60 mg%; creatinine clearance >50 - 74% | Severe albuminuria; severe hypertension; persistent anemia (<10 g%); severe renal failure; urea >60 mg%; creatinine >4 mg%; creatinine clearance <50% | Malignant hypenension;<br>uremic coma/urea<br>>100% |
| arynx-<br>ate RT Morbidity Scoring | No change from baseline | Hoarseness; slight<br>arytenoid edema | Moderate arytenoid edema; chondrids | Severe edema; severe chondritis | Necrosis |



# RTOG/EORTC Late Radiation Morbidity Scoring Scheme Use for adverse event occurring greater than 90 days after radiation therapy.

| Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| Liver-<br>Late RT Morbidity Scoring | No change from<br>baseline | Mild lassitude; nausea;<br>dyspepsia; slightly<br>abnormal liver function | Moderate symptoms:<br>some abnormal liver<br>function tests: serum<br>albumin normal | Disabling beparic insufficiency; liver function tests grossly abnormal; low alburnun; edema or ascites | Necrosis/bepotic coma or enceptual opathy |
| Lung-<br>Late RT Morbidity Scoring | No change from<br>baseline | Asymptomatic or mild symptoms (dry cough); slight radiographic appearances | Moderate symptomatic fibrosis or pneumonitis (severe cough); low grade fever; patchy radiographic appearances | Severe symptomatic<br>fibrosis or pueumonicis;<br>deuse radiographic<br>chauges | Sever respiratory in sufficiency/ continuous Oylassi sted ventilation |
| Mucous membrane-<br>Late RT Morbidity Scoring | No change from baseline | Slight atrophy and dryness | Moderate atrophy and telangiectasia: little mucus | Marked atrophy with complete dryness: severe telangiectasia | Ulcemon |
| Salivary glands-<br>Late RT Morbidity Scoring | No change from baseline | Slight dryness of mouth: good response on stimulation | Moderate dryness of mouth; poor response on stimulation | Complete drypess of mouth; no response on stimulation | Fibrosis |
| Skin-<br>Late RT Morbidity Scoring | No change from baseline | Slight atrophy;<br>pigmeatation change;<br>some hair loss | Patchy arophy;<br>moderate telangiectasia;<br>total bair loss | Marked atrophy; gross<br>telangiectasia | Ulceration |
| Small/Large intestine-<br>Late RT Morbidity Scoring | No change from<br>baseline | Mild diarrhea; mild cramping; bowel movement 5 x daily; slight rectal discharge or bleeding | Moderate diarrhes and colic; bowel movement >5 x daily; excessive rectal mucus or intermittent bleeding | Obstruction or bleeding, requiring surgery | Necrosis/perforation fistula |
| Spinal cord-<br>Late RT Morbidity Scoring | No change from baseline | Mild Lhermitte's<br>syndrome | Severe Lhermitte's syndrome | Objective neurological findings at or below cord level treatment | Moso, para-,<br>quadriplegia |
| Subcutaneous tissue-<br>Late RT Morbidity Scoring | No change from baseline | Slight induration<br>(fibrosis) and loss of<br>subcutaneous fat | Moderate fibrosis but asymptomatic: slight field costracture: <10% linear reduction | Severe induration and loss of subcutaneous tissue; field contracture >10% linear measurement | Necrosis |
| Radiation - Other<br>Specify,) | None | Mild | Moderate | Severe | Life-threatening or<br>disabling |

# BMT-Specific Adverse Events

Summary of BMT-Specific Adverse Events that may be used if specified by the protocol. These differ from the standard CTC and may be more relevant to the transplant setting. They are listed here for the convenience of investigators writing transplant protocols. They are also included in the CTC document.

| Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| Bilirubin associated with graft versus host disease for BMT studies | normal | ≥2 - <3 mg/100 mL | ≥3 - <6 mg/100 mL | ≥6 - <15 mg/100 mL<br> | ≥15 mg/100 mL |
| Diarrhea associated with graft versus host disease (GVHD) for BMT studies. | DODE | >500 - ≤1000mL of<br>diarrhea/day | >1000 · ≤1500mL of<br>diarrbea/day | > 1 500mL of<br>diarrhea/day | severe abdominal point with or without ileus |
| Diarrhea for pediatric BMT studies. | | >5 · ≤10 mL/kg uf<br>diarrhea/day | >10 · SIS mL/kg of<br>diarrhea/day | >15 mL/kg af<br>diarrheo/day | • |
| Hepatic enlargement | absent | • | • | present | _ |
| Leukocytes (total WBC) for<br>BMT studies. | WNL | ≥2.0 - <3.0 X 10° /L<br>≥2000 - <3000/mm³ | ≥1.0 - <2.0 x 10 <sup>4</sup> /L<br>≥1000 - <2000/mm <sup>3</sup> | ≥0.5 - <1.0 x 10 <sup>4</sup> /L<br>≥500 - <1000/mm³ | <0.5 x 10° /L<br><500/mm³ |
| Leukocytes (total WBC) for pediatric BMT studies (using age, race and sex normal values). | | ≥75 - <100% LLN | ≥0 · <75% LLN | ≥25 - 50% LLN | <25% ILN |
| Lymphopenia for pediatric<br>BMT studies (using age,<br>race ond sex normal values). | um, | ≥75•<100%LLN | చ0-<75%LLN | 225-<50%LLN | <25%LLN |
| Neutrophils/granulocytes<br>(ANC/AGC) for BMT<br>studies. | WNL | ≥1.0 - <1.5 x 10° /L<br>≥1000 - <1500/mm³ | ≥0.5 - <1.0 x 10° /L<br>≥500 - <1000/mm <sup>3</sup> | ≥0.1 - <0.5 x 10°/L<br>≥100 - <500/mm³ | <0.1 x 10° /L.<br><100/mm³ |
| Platelets for BMT studies. | WNL | ≥50.0 - <75.0 x 10°/L<br>≥50.000 - <75.000/mm³ | ≥20.0 - <50.0 x 10° /L<br>≥20.000 - <50.000/mm² | ≥10.0 - <20.0 x 10° /L<br>≥1u, ^0 - <20,000/mm³ | <10.0 x 10° /L<br><10,000/mm <sup>3</sup> |
| Rash/dermatitis associated with high-dose chemotherapy or BMT studies. | done . | faint erythema or dry<br>desquamation | moderate to brisk erythema or a patchy moist desquamation, mostly confined to skin folds and creases; moderate edema | confluent moist desquamation. ≥1.5 cm diameter, not confined to skin folds; pitting edema | skin accrosis or<br>ulceration of full<br>thickness dermis; may<br>include spontaneous<br>bleeding not induced b<br>minor trauma or<br>abrasion |
| Rash/desquamation associated with graft versus bost disease (GVHD) for BMT studies. | none | macular or papular eruption or erythema covering <25% of body surface area without associated symptoms | macular or papular eruption or erythema with pruritus or other associated symptoms covering 225 - <50% of body surface or localized desquamation or other lesions covering 225 - <50% of body surface area | symptomatic generalized erythroderma or symptomatic macular, papular or vesicular eruption, with bullous formation, or desquamation covering 250% of body surface area | generalized exfoliative<br>dermatitis or ulcerative<br>dermatitis or bullous<br>formation |

# BMT-Specific Adverse Events

Summary of BMT-Specific Adverse Events that may be used if specified by the protocol. These differ from the standard CTC and may be more relevant to the transplant setting. They are listed here for the convenience of investigators writing transplant protocols. They are also included in the CTC document.

| | | Gr | ade | | |
|---|---|---|---|---|---|
| Adverse Event | 0 | 1 | 2 | 3 | 4 |
| Stomatitis/pharyngins<br>(oral/pharyngeal mucositis)<br>(or BMT studies. | Botte | painless ulcers. erythema, or mild soreness in the absence of lesions | punful crythema,<br>edema or ulcers but can<br>swallow | psinful crythems, edems, or ulcers preventing swallowing or requiring hydration or parenteral (or enteral) autritional support | severe ulceration requiring prophylactic incubation or resulting in documented aspiration pneumonia |
| Transfusion: Platelets for BMT studies. | DODC | l platelet transfusion in<br>24 hours | 2 platelet transfusions (q<br>24 bours | ≥3 platelet transfusions<br>in 24 hours | platelet transfusions and other measures required to improve platelet increment; platelet transfusion refractoriness associate with life-threatening bleeding. (e.g., HLA or cross matched platelet transfusions) |
| Transfusion: pRBCs for BMT studies. | none | ≤2 u pRBC in 24 hours elective or planned | 3 u pRBC in 24 hours<br>elective or planned | ≥4 u pRBC in 24 bours | hemorrhage or<br>hemolysis associated<br>with life-threatening<br>anemia; medical<br>intervention required to<br>improve hemoglobin |
| Transfusion: pRBCs for pediatric BMT studies. | none | SI SmL/kg in 24 haurs<br>elective or planned | >15 · ≤10mL/kz in 24<br>hours elecave or<br>planned | >30mL/kg in 24 hours | hemorrhage or<br>hemolysis associated<br>with life-threatening<br>anemia; medical<br>intervention required to<br>improve h. oglobin |
| Thrombotic microangiopathy (e.g., thrombodic thrombocytopenic purpura/TTP or hemolytic uremic syndrome/HUS) for BMT studies. | - | evidence of RBC<br>destruction<br>(schistocytosis) without<br>clinical consequences | evidence of RBC destruction with elevated creatinine (S) x ULN) | evidence of RBC destruction with creatings (>3 x ULN) not requiring diatysis | evidence of RBC destruction with renal failure requiring dialysis and/or encephalopathy |
| Weight gain associated with<br>Veno-Occlusive Disease<br>(VOD) for BMT studies. | <2% | 22 - 선두 | ≥5 - <10% | ≥10% or as ascites | ≥10% or fluid recention resulting in pulmonary failure |

# ENT Complex/Multicomponent Events

| Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | | | | | |
| | 0 | 1 | 2 | 3 | 4 |
| Note: The grading of Complex/Multicomponent Events in bone marrow transplant will be defined in the protocol. The grading scale must use the CTC criteria for grading the specific component events (adverse events). | | | | | |
| Failure to engraft | absent | mld | moderate | severe | life-threatening |
| Also consider Hemoglobin, N<br>Platelets for BMT studies, if | leutrophils/granulocytes<br>specified in the protocol | (ANC/AGC), Neutrophily | granulocytes (ANC/AGC) (o | r BMT studies, if specified in | |
| Graft versus bost disease | absent | mid | moderate | severe | life-threatening |
| Also consider Fatigue, Rash/desquamation, Rash/desquamation associated with graft versus host disease (GVHD) for BMT studies, if specified in the protocol, Diarrhea for patients without colostomy. Diarrhea for patients with colostomy, Diarrhea associated with graft versus host disease (GVHD) for BMT studies, if specified in the protocol, Diarrhea for pediatric BMT studies, if specified in the protocol, Bilirubin associated with graft versus host disease (GVHD) for BMT studies, if specified in the protocol | | | | | |
| Stem cell infusion complications | absent | mild | moderate | severe | life-threatening |
| Also consider Allergic reaction/hypersensitivity, Conduction abnormality/Atrioventricular heart block, Nodal/junctional arrhythmia/dysrbythmia. Prolonged QTc interval (QTc >0.48 seconds), Sinus bradycardia. Sinus tachycardia, Supraventricular arrhythmias (SVT/atrial fibrillation/flutter), Vasovagal episode, Ventricular arrhythmia (PVCs/bigeminy/trigeminy/ventricular tachycardia), Cardiovascular/Arrhythmia - Other (Specify). Hypertension, Hypotension, Fever (in the absence of neutropenia, where neutropenia is defined as AGC <1.0 x 10°/L), Rigors/chills, Sweating (diaphoresis), Rash/desquamation, Rash/desquamation associated with graft versus host disease (GVHD) for BNT studies, if specified in the protocol, Urricaria (hives, welts, wheals), Diarrhea for patients without colostomy, Diarrhea associated with graft versus host disease (GVHD) for BMT studies, if specified in the protocol, Diarrhea for patients BMT studies, if specified in the protocol, Nausea, Vomiting, Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia, Hemorrhage/bleeding without grade 3 or 4 thrombocytopenia, Hemorrhage/bleeding without specified in the protocol, GGT, SGOT (AST), SGPT (ALT), Infection (documented clinically or microbiologically) with grade 3 or 4 neutropenia (ANC <1.0 x 10°/L), Infection without neutropenia, Hyperhaltenia, Hyperhaltenia, Depressed level of consciousness, Seizures, Abdominal pain, Hendache, Creatinine, Hemoglobinuria | | | | | |
| Veno-Occlusive Disease<br>(VOD) | absent | mild | moderate | severe | life-threatening |
| Also cons in Weight gain associated with Veno-Occlusive Disease (VOD) for BMT studies, if specified in the protocol, Bilirubia, Bilirubia associated with graft versus bost disease (GVHD) for BMT studies, if specified in the protocol, Depressed level of consciousness, Hepatic pain, Renal failure, Hepatic enlargement | | | | | |

### APPENDIX VIII

# GUIDELINES FOR REPORTING OF ADVERSE EVENTS (AE)/ ADVERSE DRUG REACTIONS (ADR) OCURRING WITH COMMERCIAL AGENTS

- 1. WITHIN 10 DAYS, SEND TO THE CITY OF HOPE IRB AND DATA SAFETY MONITORING BOARD C/O CPRMC.
- a) A COPY OF THE FDA FORM 3500
- 2. IN ADDITION, FOLLOW THE GUIDELINES BELOW

The following guidelines for reporting an AE/ADR apply to this protocol which uses commercial anticancer agents. The following AE/ADR experienced by patients accrued to this protocol and attributed to the commercial agents.

- (a) Any AE/ADR which is <u>life threatening (Grade 4)</u> or <u>fatal (Grade 5)</u> and <u>unknown</u>. Any occurrence of secondary AML or MDS must also be reported.
- (b) Any increased incidence of a known AE/ADR reported in the protocol.
- (c) Any AE/ADR which if fatal (Grade 5), even though known.<sup>3</sup>

The AE report, documented on Form FDA-3500 should be mailed to the address below within 10 working days:

or Fax to: - Medwatch 1-800-FDA-0178 5600 Fishers Lane

Rockville, MD 20852-9787

Reactions judged <u>definitely</u> not treatment related should not be reported, except that <u>all deaths</u> while on treatment or within 30 days after treatment must be reported. Any death more than 30 days after treatment which is felt to be treatment related must also be reported.

<sup>&</sup>lt;sup>1</sup> For grading reactions, see App V, VI.

<sup>&</sup>lt;sup>2</sup> All known toxicities can be found in either the drug Information, Background or in the consent form sections of the protocol.

<sup>&</sup>lt;sup>3</sup> A report shall be submitted if there is only a reasonable suspicion of drug effect.

## Appendix IX

# Eligibility Checklist #99041

# Inclusion Criteria (circle yes or No)

1. Subject has acute myelogenous or lymphocytic leukemia who are not in first remission or second remission i.e. after failing remission induction therapy or in relapse or beyond second remission, or patients with chronic myelogenous leukemia in blastic phase of the disease are eligible for the study. Patients with refractory anemia with excess blasts and in transformation will be eligible.

YES NO

Subject has a HLA (A,B,C,DR) identical siblings who is willing to donate bone
marrow for marrow grafting. All ABO blood group combinations of the
donor/recipient are acceptable since even major ABO compatibilities can be
dealt with by various techniques.

YES NO

3. A cardiac evaluation with electrocardiogram and MUGA or echocardiogram is required in all subjects and must have an ejection fracture of greater than or equal to 50%.

YES NO

4. Subject is older than 16 and the upper age limit are physiological age of 50.

YES NO

5. Subject has a serum creatinine of less than or equal to 1.2 or creatinine clearance > 80ml/min and a bilirubin of less than or equal to 1.5. Subjects should also have an SGOT and SGPT less than 5 times the upper limit of normal.

YES NO

6. The time from the last induction or reinduction attempt is greater than or equal to 28 days.

YES NO

7. Signed informed consent form approved by the IRB.

YES NO

| 8. | Pulmona | ry function tes | sts including DLCO is performed and FEV <sub>1</sub> and DLCO |
|---|---|---|---|
| | are greate | er than 50% o | f predicted normal value. |
| | | YES | NO |
| Do | nors | | |
| 9. | Is sibling | donor histoco | ompatible with the prospective recipient? |
| | | YES | NO |
| 10. | . Donor <u>do</u> e | es not have p | sychological or medical reasons and they are able to |
| | tolerate th | e procedure. | |
| - | | YES | NO |
| | | Are all | answers YES? YES NO |
| *No | te: If all ans | | circled YES then the subject is eligible to go on the study. |
| 1,500 | | | |
| Ex | clusion C | <u>riteria</u> | |
| All | answers | must be NO | (circle YES or NO) |
| 11. | Prior radia | ation therapy t | hat will exclude the use of total body irradiation. |
| | | NO | YES |
| 12. | Patients w | ho have unde | ergone bone marrow transplantation previously and |
| | who have | | |
| | | NO | YES |
| 13. | Patients w | ith psycholog | ical or medical condition that the physician deems |
| | | | d to allogeneic bone marrow transplant. |
| | | NO | YES |
| | | Are all ans | wers NO? YES NO |
| *No | te: If all ansv | vers were NO th | en the subject is eligible for study entry |
| 15.42.3 | and seems and the seems of | are lacestable are green all and a | |
| *No | te: If all the a | answers are not | YES or NO in appropriate sections then go over this case with |
| the I | Pl. If the Pl | approves an elig | ibility waiver then the reasons why must be documented in the |
| | | | arch record and a protocol deviation form must be filled out. Per |
| | | | make one waiver of the same criteria without amending the |
| stud | y and getting | g IRB approval p | rior to entry. |
| CD | Λ signatus | • | Data / / |
| | A signatur | <u> </u> | Date /_/_ |

 $i_{\omega,I}^{-s}$ 

Patient Name:

| B# 99041 (BU, FTBI, VP-16, BM<br>Eligibility Checklist | Sept. |
|---|---|
| | MR# |

| | YES | NO | DATE / RESULT |
|---|---|---|---|
| CONSENT FORM SIGNED? | IES | NO | DATE / RESULT |
| All questions must be answered "YES" to be eligible. | | \$ 34G. | |
| Patient has Acute Myelogenous Leukemia or lymphocytic | | | |
| Leukemia who is not in first remission or second remission, i.e. after failing | | | |
| remission induction therapy or in relapse or beyond second remission, or diagnosed | | } | |
| with Chronic Myelogenous Leukemia in blastic phase of the disease is eligible. | | | |
| *Patients with refractory anemia with excess blasts and in transformation will be | | ł | |
| eligible. | | | |
| 2. Patient has a HLA (A,B,C,DR) identical sibling who is willing to donate bone | | | |
| marrow for marrow grafting. (All ABO blood group combinations of the | | [ | |
| donor/recipient are acceptable ) | | | |
| 3. Ejection fraction of greater than or equal to 50%. | | | |
| 4. Patient is older than 16 and the upper age limit are physiological age of 50. | | | |
| 5. Serum Creatinine of less than or equal to 1.2 or creatinine clearance > 80 ml/min. | | | |
| 6. Bilirubin of less than or equal to 1.2 or creatinine clearance > 80 m/min. | | | |
| 7. SGOT and SGPT less than 5 times the ULN | | | |
| 8. The time of the last induction or reinduction attempt is greater than or equal to 28 | | | |
| days. | | | |
| 9. Pulmonary function tests are greater than 50% of predicted normal value. | | | |
| 10. Is the sibling donor histocompatable wit the recipient | | | |
| 11. Donor does not have psychological or medical problems and they are able to | ··· | | |
| tolerate the procedure? | | | |
| All answers must be answered "NO" to be eligible. | | 1, 7, 7, 3 | |
| 1. Prior radiation therapy that will exclude the use of total body irradiation. | | | |
| 2. The patient has undergone bone marrow transplantation previously and who have | | | |
| relapsed. | | | |
| 3. Patient with psychological or medical condition that the physician deems | | | |
| unacceptable to proceed to ALLO BMT? | | | |
| 4. Is the patient pregnant or lactating? | P.1118580408 | #137725731#F | arativi programa programa. |
| BASELINE TESTS: All testing must be completed 14 days prior to | | | |
| starting treatment. CBC, DIFF, PLT | 20 och 1985 | 1909/1919 | |
| Complete Chemistry panel | | | |
| Magnesium | | | |
| Hepatitis panel | | | |
| HIV test | | | |
| PT, PTT | | | |
| Urinalysis | | | |
| Pregnancy test | | | |
| 24 hour creatinine clearance | | | |
| CMV | | | |
| HSV/HZV | | | |
| Immunoglobulin level | | | |
| Pulmonary function test EKG | | | |
| Chest x-ray | | | |
| CT Scan of the: | | | |
| a. Chest | | - 1 | |
| b. Abdomen | | | |
| ECHO or MUGA | | | |
| Lumbar puncture (see 6.1g for conditions) | | | |
| Bone marrow: * can be done within 4 weeks* | | | |
| a. aspiration | ŀ | 1 | |
| b. biopsy | 1 | l | |
| c. cytogenetics | l | | |

| Eligibility completed by (signature & printed): |
|-------------------------------------------------|
| Date completed: |

After all eligibility has been met, fax this form, the consent form and all outside test results before the patient starts treatment

Kim Gilfillan, CCRA at City of Hope, Dept. of Biostatistics FAX: 626-256-8736 Telephone: 626-359-8111 ext. 3811

Eligibile: YES / NO **COH CRA SIGNATURE:** 

# IRB # 99041 (BU, FTBL, VP-16, BMT) Eligibility Checklist

| D 41 4 8 1 | Enginity Checkist |
|---------------|-------------------|
| Patient Name: | MR# |

| CONCENT FORM CICNODS | YES | NO | DATE / RESULT |
|---|---|---|---|
| CONSENT FORM SIGNED? | <del> </del> | <del> </del> | |
| All questions must be answered "YES" to be eligible. | 1 2.7. 0 | | FEE - 1 - 2 |
| 1. Patient has Acute Myelogenous Leukémia or lymphocytic | The state of | 133 | |
| Leukemia who is not in first remission or second remission, i.e. after failing | | | |
| remission induction therapy or in telapse or beyond second remission or diagnosed | | | 1 |
| with Chronic Myelogenous Leukemia in blastic phase of the disease is eligible. | | | |
| *Patients with refractory anemia with excess blasts and in transformation will be | | 1 | |
| eligible. | | <u> </u> | |
| 2. Patient has a HLA (A,B,C,DR) identical sibling who is willing to donate bone | 1 | 1 | |
| marrow for marrow grafting. (All ABO blood group combinations of the donor/recipient are | 1 | | |
| acceptable) | 1 | | |
| 3. Ejection fraction of greater than or equal to 50%. | <del> </del> | <del> </del> | |
| 4. Patient is older than 16 and the upper age limit are physiological age of 50. | <del> </del> | <del> </del> | |
| 5. Serum Creatinine of less than or equal to 1.2 or creatinine clearance > 80 ml/min. | <b>†</b> | † | |
| 6. Bilirubin of less than or equal to 1.5 | 1 | 1 | |
| 7. SGOT and SGPT less than 5 times the ULN | | | |
| 8. The time of the last induction or reinduction attempt is greater than or equal to 28 | | | |
| days. | <u> </u> | ļ | |
| <ol> <li>9. Pulmonary function tests are greater than 50% of predicted normal value.</li> <li>10. Is the sibling donor histocompatable wit the recipient</li> </ol> | <u> </u> | | |
| Is the storing donor histocompatable wit the recipient Donor does not have psychological or medical problems and they are able to | <del> </del> | <b></b> | |
| tolerate the procedure? | | | |
| All answers must be answered "NO" to be eligible. | - N. 1 - N. 15 | | |
| Prior radiation therapy that will exclude the use of total body irradiation. | r is the little | | |
| 2. The patient has undergone bone marrow transplantation previously and who have | <u> </u> | <del> </del> | |
| relapsed. | | | |
| 3. Patient with psychological or medical condition that the physician deems | | 1 | |
| unacceptable to proceed to ALLO BMT? | | | |
| 4. Is the patient pregnant or inctating? RASELINE TESTS: All tout | | 7. 3.5 | |
| BASELINE TESTS: All testing must be completed 14 days prior to starting treatment. | | | |
| CBC, DIFF, PLT | | <del> </del> | |
| Complete Chemistry panel | | <b> </b> | |
| Magnesium | <b></b> | | |
| Hepatitis panel | | | |
| HIV test | | | |
| PT, PIT | | | |
| Urinalysis Pregnancy test | | | |
| 24 hour creatinine clearance | | ļ | |
| CMV | | | |
| HSV/HZV | | | |
| Immunoglobulin level | | | |
| Pulmonary function test | | | |
| EKG | | | |
| Chest x-ray CT Scan of the: | | | |
| a. Chest | | | |
| b. Abdomen | | | |
| ECHO or MUGA | | | |
| Lumbar puncture (see 6.1g for conditions) | | | |
| Bone marrow: * can be done within 4 weeks* | | | |
| a. aspiration | | | |
| b. biopsy | | | |
| c. cytogenetics | | | |

| Eligibility completed by (signature & printed): | : |
|-------------------------------------------------|---|
| Date completed: | |

IRB#: 99041

### **APPENDIX X**

Time points to grade toxicities and collect data.

Day 30 after PBSCT/BMT CTC form.

Day 31 – 100 CTC form and IBMTR booklet.

101 – 365 LT Follow up form.

Every year LT follow up form.